## Statistical Analysis Plan

A Randomized Open-label Four-way Crossover Study to Compare the Pharmacokinetics, Safety, and Tolerability of Three Different Formulations of M207 3.8 mg (Administered as two 1.9 mg patches) on the Upper arm for 30 Minutes with Intranasal Zolmitriptan 2.5 mg in Healthy Volunteers

Protocol No: CP-2019-002
Final Protocol Date: 15 April 2019

Protocol Clarification Letter 1: 18 April 2019 Protocol Clarification Letter 2: 23 May 2019

Compound Name: M207 (Zolmitriptan Microneedle System)

Celerion Project CA27752 Final Version Date: 04 July 2019

Zosano Pharma Corporation 34790 Ardentech Court Fremont, CA 94555, United States

Celerion 100 Alexis-Nihon Boulevard, Suite 360 Montreal, QC, H4M 2N8, Canada

## Statistical Analysis Plan Signature Page

| ! | |
|---|---|
| Compound Name: M207 (Zolmitriptan Microneedle Sy | ystem) |
| Protocol: CP-2019-002 | |
| Study Title: A Randomized Open-label Four-way Cros Pharmacokinetics, Safety, and Tolerability of Three Di (Administered as two 1.9 mg patches) on the Upper arm Zolmitriptan 2.5 mg in Healthy Volunteers | fferent Formulations of M207 3.8 mg |
| Issue Date: 04 July 2019 Tamas Civild<br>Director, Biss | hy<br>Hadistics |
| Signature Sangar Olarly<br>deligate for Sanyath Radji, MSc | Date: 10 Jul 2019 |
| Biostatistician II, Data Management and Bio | ometrics |
| Celerion<br>100 Alexis-Nihon Boulevard, Suite 360 | |
| Montreal, QC H4M 2N8, Canada | |
| Signature: 1. Moulin | Date: 10-JUL-2019 |
| Ted Marenco, MSc Senior Pharmacokineticist II, | |
| Clinical Pharmacology and Pharmacometric | 58, |
| Data Management and Biometrics Celerion | |
| 100 Alexis-Nihon Boulevard, Suite 360 | |
| Montreal, QC II4M 2N8, Canada | |
| Signature: January for Lold | Date 7-07-2019 |
| Don Kellerman VP, Clinical Development and Regulatory A | |
| Zosano Pharma Corporation | 1110113 |
| Signature: 1. S. | Date: 7/5/2019 |
| Izan M. Engels, MS | |
| Director, Biostatistics | |
| Zosano Pharma Corporation | |

## **Table of Contents**

| 1. | INT. | RODUCTION | 5 |
|---|---|---|---|
| 2. | OBJ | ECTIVES AND ENDPOINTS | 5 |
| | 2.1 | Objectives | |
| | 2.2 | Endpoints | |
| 3. | STU | DY DESIGN | . 6 |
| | | ALYSIS POPULATIONS | |
| 4. | | | |
| | 4.1<br>4.2 | Analysis PopulationsPreliminary Analysis of Pharmacokinetic Data | |
| _ | | | |
| 5. | | ATMENT DESCRIPTIONS | |
| 6. | PHA | RMACOKINETIC ANALYSIS | |
| | 6.1 | Measurements and Collection Schedule | |
| | 6.2 | Bioanalytical Method | 9 |
| | | 6.2.1 Plasma Zolmitriptan | 9 |
| | | 6.2.2 Plasma N-Desmethyl Zolmitriptan | 9 |
| | | 6.2.3 Residual Zolmitriptan in Patches and Skin Swabs | 9 |
| | 6.3 | Investigational Product and PK Analyte Information | |
| | | 6.3.1 Zolmitriptan | 9 |
| | | 6.3.2 N-Desmethyl Zolmitriptan | 10 |
| | 6.4 | Pharmacokinetic Concentrations | |
| | 6.5 | NonCompartmental Pharmacokinetic Analysis and Parameter Calculation | 10 |
| | 6.6 | Data Summarization and Presentation | |
| | 6.7 | Statistical Analysis of PK Parameters | 13 |
| 7. | SAF | ETY | 14 |
| , | 7.1 | Subject Discontinuation | |
| | 7.2 | Demographics | |
| | 7.3 | Adverse Events | |
| | 7.4 | Clinical Laboratory Tests | 15 |
| | 7.5 | Vital Signs | 16 |
| | 7.6 | Electrocardiogram | 16 |
| | 7.7 | Concomitant Medications | 17 |
| | 7.8 | Physical Examination | |
| | 7.9 | Investigator Visual Skin Assessment | 17 |
| 8. | SUN | IMARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS | 18 |
| 9. | SUM | IMARY TABLES AND FIGURES | 18 |
| | 9.1 | In-text Summary Tables and Figures | 19 |
| | 9.2 | Section 14 Summary Tables and Figures | 20 |

## Zosano Pharma Corporation M207, CP-2019-002 Celerion, Clinical Study Report No. CA27752

| | 9.3 | Section 16 Data Listings | 25 |
|-----|------|----------------------------------|----|
| 10. | | LE AND FIGURE SHELLS | |
| | | In-text Summary Tables Shells | |
| | | Figures Shells | |
| | | Section 14 Summary Tables Shells | |
| 11. | LIST | ING SHELLS | 61 |

#### 1. INTRODUCTION

The following statistical analysis plan (SAP) provides the framework for the summarization of the data from this study. The SAP may change due to unforeseen circumstances. Any changes made from the planned analysis within the protocol, after the locking of the database will be documented in the clinical study report CSR. The section referred to as Table Shells within this SAP describes the traceability of the tables, figures, and listings (TFLs) back to the data. Note that the header for this page will be the one used for the main body of the CSR.

Any additional exploratory analyses not addressed within this statistical analysis plan (SAP) and/or driven by the data, or requested by Zosano Pharma Corporation, will be considered out of scope and must be described in the CSR.

### 2. OBJECTIVES AND ENDPOINTS

## 2.1 Objectives

- To compare the pharmacokinetics (PK), safety and tolerability of M207 3.8 mg (Sled) (Treatment A) to M207 3.8 mg (MACAP) (Treatment B) to M207 3.8 mg (MiniMac) (Treatment C), each worn for 30 minutes on the upper arm.
- To compare the PK, safety and tolerability of these 3 formulations of M207 3.8 mg to intranasal zolmitriptan 2.5 mg (Treatment D).

### 2.2 Endpoints

### Safety and Tolerability

- · Incidence of adverse events
- Change in physical exam findings from predose to 8 hr postdose
- Changes in vital signs from predose to 10 minutes, 60 minutes, and 2, 4 and 12 hr postdose
- Changes in ECG parameters from predose to 15 minutes and 12 hr postdose
- Scores from the investigator's visual skin assessment for erythema, edema, bruising and bleeding at the patch application sites from predose to 30 minutes, 60 minutes, 8 hr and 24 hr postdose

## Pharmacokinetics

- Cmax maximum observed plasma concentrations
- Tmax time to maximum concentration
- AUC0-t the area under the plasma concentration time profile from hour 0 to the last detectable concentration at time t.
- AUC0-30min the area under the plasma concentration time profile from minute 0 to minute 30.
- AUC0-60min the area under the plasma concentration time profile from minute 0 to minute 60.
- AUC0-120min the area under the plasma concentration time profile from minute 0 to minute 120
- Kel apparent elimination rate constant will be estimated by linear regression of the log-transformed plasma concentrations during the terminal log-linear decline phase.
- $t\frac{1}{2}$  apparent half-life ( $t\frac{1}{2}$ ) values will be calculated as 0.693/Kel.
- AUC0-inf the AUC value extrapolated to infinity will be calculated as the sum of AUC0-t, and the area extrapolated to infinity, calculated by the concentration at time t (Ct) divided by k.
- AUC0-inf(m/p) metabolite to parent ratio of AUC0-inf
- %Frel bioavailability relative to each treatment assignment

#### 3. STUDY DESIGN

This is a single-center, open-label, randomized, four-way crossover study. The study population will consist of 24 healthy volunteers (12 women and 12 men) 18 to 50 years of age in general good health. Following review of all Screening procedures, eligible subjects will be enrolled into the dosing phase of the study. The interval between screening and first treatment will be no more than 30 days.

Eligible subjects will be admitted into the clinic on the day before the first dosing. Subjects will be required to stay in the clinic for the entire duration of the study (unless medically necessary to leave the clinic as instructed by the principal investigator and/or for non-medically related reasons considered on a case by case basis).

Subjects will fast for at least 10 hours during the night preceding dosing and until at least 2 hours after dosing. Water is allowed ad libitum, as well as tea and coffee in moderate amounts. The following morning (between 0630 and 0930), subjects will receive that day's scheduled treatment (A, B, C, or D). The treatments are described in Section 5. Hour 0 will be the time of second patch application.

Each subject will receive each of the 4 study treatments once, followed by in-clinic monitoring and extensive blood sample collections for PK analysis. All AEs,

including any skin irritations and sensations as well as concomitant medication usage will be documented.

Depending on the treatment assignment, two M207 patches (Treatments A, B, and C) will be applied to the upper arm by means of a handheld reusable applicator with an application energy of 0.26 Joules. No lotions, ointments, or powders may be applied to the upper arm where M207 will be applied for 12 hours before or after applying M207. Used patches will be removed 30 minutes after application of the second patch. The patches will be collected and frozen in storage until shipped for analysis of remaining drug. For Treatment D (nasal spray), the dose will be administered, after the subject blows his/her nose, to either the right or left nostril with the subject's head tilted slightly backward.

Dosing will occur approximately 48 hours apart from the time of patch application, until completion of dosing in randomized order per the treatment sequence schedule. Treatments sequences ABDC, BCAD, CDBA, and DACB will be used. At the end of each dosing day, the safety data from the subjects will be evaluated. If tolerability is deemed to be acceptable by the Principal Investigator, a decision will be made to proceed to the next dosing day. After completion of the four dosing days (one in each treatment period), subjects will be assessed one final time and dismissed from the study.

## 4. ANALYSIS POPULATIONS

## 4.1 Analysis Populations

## **Safety Population**

The safety population will include all subjects who received any amount of study drug.

#### Pharmacokinetic Population

The PK population will include all subjects who were dosed and who have an evaluable PK profile.

## 4.2 Preliminary Analysis of Pharmacokinetic Data

Celerion will perform a preliminary analysis of plasma zolmitriptan and n-desmethyl zolmitriptan PK data. PK parameters will be calculated using quality-controlled plasma zolmitriptan and n-desmethyl zolmitriptan concentration data and actual sampling times.

## 5. TREATMENT DESCRIPTIONS

The treatments descriptions will be described as:

| Treatment | Short Description | Long Description |
|---|---|---|
| Treatment A | M207 3.8 mg (Sled) | M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "Sled" coater and packaged in foil pouches (Treatment A) |
| Treatment B | M207 3.8 mg (MACAP) | M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "MACAP" coater and packaged in foil cups (Treatment B) |
| Treatment C | M207 3.8 mg (MiniMac) | M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "MiniMac" coater and packaged in foil cups (Treatment C) |
| Treatment D | Zolmitriptan 2.5 mg (Intranasal) | Zolmitriptan 2.5 mg administered intranasally as a single 2.5 mg/0.1 mL spray (Treatment D) |

## 6. PHARMACOKINETIC ANALYSIS

## 6.1 Measurements and Collection Schedule

Blood samples for the determination of plasma zolmitriptan and n-desmethyl zolmitriptan concentrations will be collected predose and 0.0333 (2 minutes), 0.0833 (5 minutes), 0.1667 (10 minutes), 0.25 (15 minutes), 0.3333 (20 minutes), 0.5 (30 minutes), 0.75 (45 minutes), 1, 1.5, 2, 4, 8, 12, and 24 hours postdose.

Following removal of the patches 30 minutes postdose, the subjects' skin will be swabbed and both the patches and skin swabs will be analyzed for residual zolmitriptan.

All plasma concentration data will be included in the calculation of the individual PK parameters, the individual concentration-time plots (based on actual sample times), and in the mean concentration-time plots (based on nominal sample times). All deviations and excluded data will be provided and discussed in the CSR.

## 6.2 Bioanalytical Method

## 6.2.1 Plasma Zolmitriptan

Plasma concentrations of zolmitriptan will be determined using a high performance liquid chromatography-tandem mass spectrometry (HPLC-MS/MS) method validated with respect to accuracy, precision, linearity, sensitivity, and specificity at Syneos Health. The analytical range (lower limit of quantitation [LLOQ] – upper limit of quantitation [ULOQ]) for zolmitriptan in plasma is expected to be 100 to 20000 pg/mL.

## 6.2.2 Plasma N-Desmethyl Zolmitriptan

Plasma concentrations of n-desmethyl zolmitriptan will be determined using a HPLC-MS/MS method validated with respect to accuracy, precision, linearity, sensitivity, and specificity at Syneos Health. The analytical range for n-desmethyl zolmitriptan in plasma is expected to be 50 to 10000 pg/mL.

## 6.2.3 Residual Zolmitriptan in Patches and Skin Swabs

Residual amounts of zolmitriptan in patches and skin swabs will be determined using HPLC-MS/MS methods validated with respect to accuracy, precision, linearity, sensitivity, and specificity at Syneos Health. The analytical range for zolmitriptan in patches and skin swabs is expected to be 7.5 to 1500 µg.

## 6.3 Investigational Product and PK Analyte Information

### 6.3.1 Zolmitriptan

Plasma will be analyzed for zolmitriptan concentrations. The analyte can be described with the following structure and molecular weight (MW) of 287.36 g/mol (Figure A). Zolmitriptan will be administered transdermally to subjects in 3.8 mg doses via Zosana M207 (Zolmitriptan Microneedle System) patches (2 patches x 1.9 mg/patch) made from 3 different types of equipment, and intranasally via a commercially available nasal spray (Zomig<sup>®</sup> Nasal Spray) at a dose of 2.5 mg (0.1 mL spray x 2.5 mg/0.1 mL).

Figure A: Zolmitriptan (MW = 287.36 g/mol)

## 6.3.2 N-Desmethyl Zolmitriptan

Plasma will be analyzed for n-desmethyl zolmitriptan concentrations. The analyte can be described with the following structure and molecular weight (MW) of 273.34 g/mol (Figure B).

Figure B: N-Desmethyl Zolmitriptan (MW = 273.34 g/mol)

## 6.4 Pharmacokinetic Concentrations

Plasma concentrations of zolmitriptan and n-desmethyl zolmitriptan as determined at the collection times and per the bioanalytical method described in Section 6.1 and Section 6.2, respectively, will be used for the calculation of the plasma zolmitriptan and n-desmethyl zolmitriptan PK parameters.

## 6.5 NonCompartmental Pharmacokinetic Analysis and Parameter Calculation

The appropriate noncompartmental PK parameters will be calculated from the plasma zolmitriptan and n-desmethyl zolmitriptan concentration-time data using Phoenix® WinNonlin® Version 7.0 or higher. Actual sample times will be used in the calculations of the PK parameters. The calculation of the actual times will be in respect to the start of patch administration (Treatments A, B, and C) or in respect to the start time of intranasal administration (Treatment D) of zolmitriptan on Day 1. All PK parameters included in the protocol are listed in Table 6.1 below, and are defined as appropriate for study design.

Table 6.1. Noncompartmental Pharmacokinetic Parameters to be Calculated

| Label to be Used in the Text, Tables and Figures Cmax Cmax | | Definition | Method of Determination Taken directly from bioanalytical data |
|---|---|---|---|
| | | Maximum observed plasma concentrations | |
| Tmax | Tmax | Time to maximum concentration | Taken from clinical database as the difference in the time of administration and the time of the blood draw which is associated with the Cmax. |
| AUC0-last AUC0-t | | Area under the plasma concentration-time profile from hour 0 to the last detectable concentration at time t | Calculated using the Linear Trapezoidal with Linear Interpolation Method |
| AUC0-30min | AUC0-30min | Area under the plasma concentration-time profile from minute 0 to minute 30 | Calculated using the Linear Trapezoidal with Linear Interpolation Method |
| AUC0-60min AUC0-60min I | | Area under the plasma concentration-time profile from minute 0 to minute 60 | Calculated using the Linear Trapezoidal with Linear Interpolation Method |
| - ( | | Area under the plasma concentration-time profile from minute 0 to minute 120 | Calculated using the Linear Trapezoidal with Linear Interpolation Method |
| k Kel | | Apparent elimination rate constant | Estimated by linear regression of the log-transformed plasma concentrations during the terminal log-linear decline phase |
| t1/2 | t½ | Apparent half-life | Calculated as 0.693/Kel |
| pl<br>cc<br>cc<br>ex | | Area under the plasma concentration-time curve from minute 0 extrapolated to infinity | Calculated as AUC0-t + (Clast/Kel) where Clast is the last observed/measured concentration |
| ratio of th<br>under the<br>concentra<br>curve froi<br>extrapola<br>infinity | | Metabolite to parent<br>ratio of the area<br>under the plasma<br>concentration-time<br>curve from minute 0<br>extrapolated to<br>infinity | Calculated as AUC0-inf of n-desmethyl zolmitriptan x (molecular weight of zolmitriptan/molecular weight of n-desmethyl zolmitriptan)/AUC0-inf of zolmitriptan, where the molecular weights of zolmitriptan and n-desmethyl zolmitriptan are 287.36 g/mol and 273.34 g/mol, respectively. |
| Frel %Frel Relative bioavailability only) | | | Bioavailability relative to each treatment assignment will be calculated as follows: %Frel(A/B) = AUC0-inf(A)/AUC0-inf(B)x100 %Frel(A/C) = AUC0-inf(A)/AUC0-inf(C)x100 %Frel(A/D) = [AUC0-inf(A)/Dose(A)]/[AUC0-inf(D)/Dose(D)]x100 %Frel(B/C) = AUC0-inf(B)/AUC0-inf(C)x100 %Frel(B/D) = [AUC0-inf(B)/Dose(B)]/[AUC0-inf(D)/Dose(D)]x100 %Frel(C/D) = [AUC0-inf(C)/Dose(C)]/[AUC0-inf(D)/Dose(D)]x100 |

For the calculation of the PK parameters, plasma zolmitriptan and n-desmethyl zolmitriptan concentrations below the limit of quantitation (BLQ) prior to the first quantifiable concentration will be set to 0.00 and plasma concentrations BLQ after the first quantifiable concentration will be treated as missing.

Pharmacokinetic parameters will not be calculated for subjects with less than 3 consecutive postdose time points with quantifiable concentrations. Subjects for whom there are insufficient data to calculate the PK parameters will be included in the concentration tables only.

For Treatments A, B, and C, subjects for whom one or both patches detach either partially or completely prior to the completion of the 30 minute wear time may be excluded from any statistics. For Treatment D, subjects who vomit or who experience nasal drip within twice the median Tmax value of 3 hours for the study drug, i.e., within first 6 hours postdose, may be excluded from any statistics.

The Kel will be determined using linear regressions composed of least 3 data points. The Kel will not be assigned if 1) the terminal elimination phase is not apparent, 2) if Tmax is one of the 3 last data points, or 3) if the R<sup>2</sup> value is less than 0.75. In cases where the Kel interval is not assigned, the values of any AUC requiring Kel for extrapolation, t½, AUC0-inf, AUC0-inf(m/p), and %Frel are considered not calculable and will not be reported. Wherever the resulting t½ is more than half as long as the sampling interval, the Kel values and associated parameters (any AUC requiring Kel for extrapolation, t½, AUC0-inf, AUC0-inf(m/p), and %Frel) may not be presented as judged appropriate and in accordance with Celerion SOPs.

The nominal doses of Treatments A, B, and C (3.8 mg), and Treatment D (2.5 mg) will be used in the calculation of the different %Frel parameters.

### 6.6 Data Summarization and Presentation

For the preliminary PK analysis, all zolmitriptan and n-desmethyl zolmitriptan PK concentrations and/or PK parameter descriptive statistics will be generated using Phoenix® WinNonlin® Version 7.0 or higher. For the final PK analysis, all zolmitriptan and n-desmethyl zolmitriptan PK concentrations and/or PK parameter descriptive statistics will be generated using SAS® Version 9.3 or higher.

The plasma concentrations of zolmitriptan and n-desmethyl zolmitriptan will be listed and summarized by treatment and time point for all subjects in the PK Population. Plasma concentrations of zolmitriptan and n-desmethyl zolmitriptan will be presented with the same level of precision as received from the bioanalytical laboratory. Summary statistics, including sample size (n), arithmetic mean (Mean), standard deviation (SD), coefficient of variation (CV%), standard error of the mean (SEM), minimum, median, and maximum will be calculated for all nominal concentration time points Excluded subjects will be included in the concentration listings, but will be excluded from the summary statistics and noted as such in the tables. All BLQ

values will be presented as "BLQ" in the concentration listings and footnoted accordingly.

The residual amounts of zolmitriptan in each patch and on the skin surface beneath each patch will be listed and the residual amounts of zolmitriptan in both patches combined and on the skin surfaces under both patches combined will be summarized by treatment for all subjects in the PK Population. Residual amounts of zolmitriptan that are BLQ will be set to 0.00. Residual amounts of zolmitriptan in patches and skin swabs will be presented with the same level of precision as received from the bioanalytical laboratory. Summary statistics, including sample size (n), arithmetic mean (Mean), standard deviation (SD), coefficient of variation (CV%), standard error of the mean (SEM), minimum, median, and maximum will be calculated for residual amounts of zolmitriptan in both patches combined and on the skin surfaces under both patches combined. Excluded subjects will be included in the listings, but will be excluded from the summary statistics and noted as such in the tables. All BLQ values will be presented as "BLQ" in the listings and footnoted accordingly.

Mean and individual plasma concentration-time profiles will be presented on linear and semi-log scales. Linear mean plots will be presented with and without SD.

Plasma zolmitriptan and n-desmethyl zolmitriptan PK parameters will be listed and summarized by treatment for all subjects in the PK Population. Pharmacokinetic parameters will be reported to 3 significant figures for individual parameters, with the exception of Tmax, which will be presented with 2 decimal places. Summary statistics (n, Mean, SD, CV%, SEM, minimum, median, maximum, geometric mean (Geom Mean), and geometric CV% (Geom CV%)) will be calculated for plasma zolmitriptan and n-desmethyl zolmitriptan PK parameters. Excluded subjects will be listed in the PK parameter tables, but will be excluded from the summary statistics and noted as such in the tables.

The level of precision for each concentration and PK parameter statistic will be presented as follows: minimum/maximum in same precision as in bioanalytical data and/or parameter output, mean/median/geometric mean in one more level of precision than minimum/maximum, SD/SEM in one more level of precision than mean/median/geometric mean, n will be presented as an integer, and CV%/geometric CV% will be presented to the nearest tenth.

## 6.7 Statistical Analysis of PK Parameters

No inferential statistics will be performed on the PK data from this study.

#### 7. SAFETY

All case report form (CRF) data will be listed by subject and chronologically by assessment time points. This will include rechecks, unscheduled assessments, and early termination.

Applicable continuous variables will be summarized using n, arithmetic mean, SD, minimum, median, and maximum.

The level of precision will be presented as follows: minimum/maximum in the same precision as in the database, mean/median in one more precision level than minimum/maximum, SD in one more precision level than mean/median, and n will be presented as an integer.

Where individual data points are missing because of dropouts or other reasons, the data will be summarized based on reduced denominators.

No inferential statistics will be performed for safety assessments.

## 7.1 Subject Disposition

Subjects will be summarized by number of subjects enrolled (randomized), completed, and discontinued the study with discontinuation reasons by randomized treatment sequence and overall. The number of subjects in the safety population will also be summarized. The individual subject's dosing status will also be provided along with their completion status and date of study completion.

## 7.2 Demographics

Descriptive statistics will be calculated for continuous variables (age, weight, height, and body mass index [BMI]) by randomized treatment sequence and overall. Weight, height and BMI will be summarized at screening. Age will be derived from date of birth to date of informed consent. Frequency counts will be provided for categorical variables (race, ethnicity, and sex) for each randomized treatment sequence and overall.

#### 7.3 Adverse Events

All adverse events (AEs) occurring during this clinical trial will be coded using the Medical Dictionary for Regulatory Activities (MedDRA®), Version 20.1.

Each AE will be graded on a 3-point severity scale (mild, moderate, severe). Similarly, the causal relationship of the study drug to the AE will be described using a 3-point relationship scale (probably related, possibly related, not related). All AEs captured in the database will be listed in by-subject data listings including verbatim term, coded term, treatment, severity, relationship to study medication, and action; however, only treatment-emergent AEs (TEAEs) will be summarized.

A TEAE is defined as an AE that is starting or worsening at the time of or after study drug administration. Each TEAE will be attributed to a treatment based on the onset date and time of the AE. An AE that occurs during the washout period between drugs will be considered treatment-emergent to the last drug administered prior to onset of the AE.

If the onset time of an AE is missing and the onset date is the same as the treatment dosing date, then the AE will be considered treatment emergent in the current treatment. If onset time of an AE is missing and the onset date does not fall on a dosing date, then the AE will be considered treatment emergent for the last treatment administered. If the onset date of an AE is missing, then the AE will be considered treatment emergent and attributed to each treatment on the study, unless the onset date is known to have occurred within or between specific treatment periods or otherwise specified.

TEAEs will be tabulated by System Organ Class (SOC) and Preferred Term. Summary tables will include number of subjects reporting the AE and as percent of number of subjects dosed by treatment. The number of AEs will be tabulated in a similar manner. Tables which tabulate the number of TEAEs by severity and relationship to study drug will also be included.

Serious adverse events (SAEs), if present, will also be listed. Applicable narratives will be included in the CSR.

## 7.4 Clinical Laboratory Tests

Standard clinical laboratory tests (chemistry, hematology, urinalysis, and serum pregnancy for all women) will be performed at Screening and End of Study (EOS, Day 3 of Period 4) or upon early termination. A serum pregnancy test will also be completed for all women on Day -1 of Period 1. Urine drug screen and alcohol testing will be performed at Screening and on Day -1 of Period 1. Screening serological tests for HIV, Hepatitis B and Hepatitis C will be performed. All clinical laboratory test results will be presented in by-subject data listings.

Out-of-normal range flags will be recorded as follows: high (H) and low (L) for numerical results and did-not-match (\*) for categorical results. If a value fails the reference range, it will automatically be compared to a computer clinically significant (CS) range. If the value falls within the computer CS range, it will be noted as "N" for not clinically significant. If the value fails (i.e., fall outside of the CS range) the computer CS range, it will be flagged with a "Y" which prompts the PI to determine how the out-of-range value should be followed using 4 Investigator flags: "N", not clinically significant, "R", requesting a recheck, "^", checking at the next scheduled visit, or "Y", clinically significant. To distinguish the PI flag from the computer CS range flags, the PI flags of "N" and "Y" will be presented as "-" and "+", respectively, in the data listing. Additionally, the PI will provide a 4th flag when the

 $3^{rd}$  flag indicates "R" or "^". This  $4^{th}$  flag is intended to capture final CS (+)/NCS (-) when the  $3^{rd}$  flag does not document significance.

Out-of-range serum chemistry, hematology and urinalysis values and corresponding recheck results will be listed. Results that are indicated as CS by the PI (in either PI flag) will be listed in a table.

## 7.5 Vital Signs

Single measurements of body temperature, respiratory rate, blood pressure (systolic and diastolic), and pulse rate will be performed at the following time points:

**Table 7.1. Vital Signs Collection Time Points** 

| Period | Day | Time Point |
|------------|---------------------|-------------------------------------|
| Screen | | |
| 1004 | -1** | |
| 1, 2, 3, 4 | 1 | Predose, 10 min, 60 min, 2 hours, 4 |
| | | hours, and 12 hours postdose |
| 4 | 3 | End of Study or Early Termination |
| | Screen 1, 2, 3, 4 4 | Screen 1, 2, 3, 4 -1** 1 |

<sup>\*</sup> Temperature will only be collected at screening, on Day -1 of Period 1, and End of Study of upon early termination.

\*\* Period 1 only

All vital signs data will be listed by subject. Descriptive statistics will be reported for vital signs parameters, excluding temperature, by treatment and assessment time point. Change from baseline will be summarized in a similar manner. Baseline will be defined as the result closest and prior to dosing in each period, including unscheduled or recheck results, whichever is later. This will typically be the predose measurement collected on Day 1 prior to dosing. Change from baseline will not be calculated for the End of Study time point. Postdose unscheduled events or rechecks will not be included in summaries. Similarly, early termination results will not be included in summaries.

## 7.6 Electrocardiogram

Safety 12-Lead ECG parameters (i.e., HR, PR, QRS, QT, and QTcF [QT corrected for heart rate using Fridericia's equation]) will be measured at the following time points:

Table 7.2. Safety 12-lead ECG Collection Time Points

| ECG Parameter | Period | Day | Time Point |
|---|---|---|---|
| | Screen | | |
| HR, PR, QRS, QT,<br>QTcF | 1, 2, 3, 4 | 1 | Predose, 15 min, and 12 hours postdose |

| ECG Parameter | Period | Day | Time Point |
|---------------|--------|-----|-----------------------------------|
| | 4 | 3 | End of Study or Early Termination |

All ECG parameters will be listed by subject and time point of collection with QTcF > 450 msec and change from baseline > 30 msec flagged. Descriptive statistics will be reported for ECG parameters by treatment and assessment time point. Change from baseline will be summarized in a similar manner. Baseline will be defined as the result closest and prior to dosing in each treatment period, including unscheduled or recheck results, whichever is later. This will typically be the predose measurement collected on Day 1 prior to dosing. Change from baseline will not be calculated for the End of Study time point. Postdose unscheduled events or rechecks will not be included in summaries. Similarly, early termination results will not be included in summaries.

## 7.7 Concomitant Medications

All concomitant medications recorded during the study will be coded with the WHO Dictionary Version 01Mar2019-b3 and listed.

## 7.8 Physical Examination

Physical examinations will be performed at Screening and 8 hours postdose in each period and EOS (Day 3 of Period 4). Abnormal findings will be reported as medical history or adverse events. All abnormal findings will be listed.

## 7.9 Investigator Visual Skin Assessment

Each M207 patch site (where a patch has been removed) will be observed by the investigator for erythema, edema, bruising, and bleeding assessments at the following time points:

Table 7.3. Investigator Visual Skin Assessment Time Points

| Skin Assessment | Period* | Day | Time Point |
|---|---|---|---|
| Erythema, Edema,<br>Bruising, Bleeding | 1, 2, 3, 4 | 1 | Predose, 30 min, 60 min, 8 hours, and 24 hours postdose |

<sup>\*</sup> The skin assessments will be performed at the specified time points for Treatments A, B, C. The predose assessment will also be performed prior to Treatment D dosing.

The erythema evaluations will be performed using the following scale:

- 0 = None
- 1 = Mild redness
- 2 = Moderate colored redness

#### 3 =Beet colored redness

The edema evaluations will be performed using the following scale:

- 0 = None
- 1 = Slight edema
- 2 = Moderate edema
- 3 =Severe edema

Bruising assessments (visual rating) will be performed using the following scale:

- 0 = None
- $1 = \le 25\%$  application site has bruising spots
- $2 = \ge 26$  to  $\le 50\%$  application site has bruising spots
- 3 = > 50% application site has bruising spots

Bleeding will be assessed using the following scale:

- 0 = None
- 1 = Pink color on skin
- 2 = Visible blood drop
- 3 = Active bleeding

Scales from the investigator skin assessment of the application sites will be listed by subject and summarized. For each treatment period, assessments will be performed for each patch application site, separately. For the purpose of the analysis, the worst scale between the two patches at each treatment will be used in the summary statistics. For each type of assessment, frequency counts and percentages showing the number of subjects obtaining each scale by treatment and time point will be provided. Percentages will be based on the number of non-missing results per treatment and time point. Descriptive statistics will also be provided for each type of assessment scales by treatment and time point. The average scale for each assessment will be plotted against time.

## 8. SUMMARY OF CHANGES FROM PROTOCOL-PLANNED ANALYSIS

The analyses described in this SAP are aligned with those analyses described in the protocol.

## 9. SUMMARY TABLES AND FIGURES

Summary tables and figures are numbered following the International Conference on Harmonization (ICH) structure but may be renumbered as appropriate during the compilation of the tables and figures for the CSR. Note that all summary tables and figures will be generated using SAS® Version 9.3 or higher and/or using Phoenix® WinNonlin® Version 6.3 or higher, as appropriate.

## 9.1 In-text Summary Tables and Figures

The following is a list of table and figure titles that will be included in the text of the CSR. Tables and figures will be numbered appropriately during compilation of the CSR.

## Section 10:

Table 10-1 Subject Disposition Summary

### Section 11:

- Table 11-1 Demographic Summary
- Figure 11-1 Arithmetic Mean (SD) Plasma Zolmitriptan Concentration-Time
  Profiles for 3 Different Formulations of M207 3.8 mg on the Upper
  Arm for 30 Minutes and Intranasal Zolmitriptan 2.5 mg in Healthy
  Volunteers (Predose to 24 Hours Postdose)
- Figure 11-2 Arithmetic Mean (SD) Plasma Zolmitriptan Concentration-Time Profiles for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes and Intranasal Zolmitriptan 2.5 mg in Healthy Volunteers (Predose to 2 Hours Postdose)
- Table 11-2 Summary of Plasma Zolmitriptan Pharmacokinetics for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes and Intranasal Zolmitriptan 2.5 mg in Healthy Volunteers
- Table 11-3 Relative Bioavailability Between Each Treatment for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes and Intranasal Zolmitriptan 2.5 mg in Healthy Volunteers
- Table 11-4 Residual Amounts of Zolmitriptan in M207 Patches and on Skin Swabs for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes in Healthy Volunteers
- Figure 11-3 Arithmetic Mean (SD) Plasma N-Desmethyl Zolmitriptan
  Concentration-Time Profiles for 3 Different Formulations of M207
  3.8 mg on the Upper Arm for 30 Minutes and Intranasal Zolmitriptan
  2.5 mg in Healthy Volunteers

## Section 12:

- Table 12-1 Treatment-Emergent Adverse Event Frequency by Treatment- Number of Subjects Reporting the Event (% of Subjects Dosed)
- Figure 12-1 Mean Investigator Visual Erythema Assessment Scale by Time Profile

- Figure 12-2 Mean Investigator Visual Edema Assessment Scale by Time Profile
- Figure 12-3 Mean Investigator Visual Bruising Assessment Scale by Time Profile
- Figure 12-4 Mean Investigator Visual Bleeding Assessment Scale by Time Profile

## 9.2 Section 14 Summary Tables and Figures

The following is a list of table and figure titles that will be included in Section 14 of the report. Table and figure titles may be renumbered as appropriate during the compilation of the report.

## 14.1 Demographic Data Summary Tables

- Table 14.1.1 Summary of Disposition (All Randomized Subjects)
- Table 14.1.2 Subject Dosing Status and Study Disposition (Safety Population)
- Table 14.1.3 Demographic Summary (Safety Population)

## 14.2 Pharmacokinetic Data Summary Tables and Figures

## 14.2.1 Plasma Zolmitriptan Tables

- Table 14.2.1.1 Plasma Zolmitriptan Concentrations (pg/mL) for M207
  3.8 mg (Sled) on the Upper Arm for 30 Minutes in Healthy
  Volunteers (Treatment A) (Pharmacokinetic Population)
- Table 14.2.1.2 Plasma Zolmitriptan Concentrations (pg/mL) for M207 3.8 mg (MACAP) on the Upper Arm for 30 Minutes in Healthy Volunteers (Treatment B) (Pharmacokinetic Population)
- Table 14.2.1.3 Plasma Zolmitriptan Concentrations (pg/mL) for M207 3.8 mg (MiniMac) on the Upper Arm for 30 Minutes in Healthy Volunteers (Treatment C) (Pharmacokinetic Population)
- Table 14.2.1.4 Plasma Zolmitriptan Concentrations (pg/mL) for Intranasal Zolmitriptan 2.5 mg in Healthy Volunteers (Treatment D) (Pharmacokinetic Population)
- Table 14.2.1.5 Plasma Zolmitriptan Pharmacokinetic Parameters for M207 3.8 mg (Sled) on the Upper Arm for 30 Minutes in Healthy Volunteers (Treatment A) (Pharmacokinetic Population)
- Table 14.2.1.6 Plasma Zolmitriptan Pharmacokinetic Parameters for M207 3.8 mg (MACAP) on the Upper Arm for 30 Minutes in Healthy Volunteers (Treatment B) (Pharmacokinetic Population)

- Table 14.2.1.7 Plasma Zolmitriptan Pharmacokinetic Parameters for M207 3.8 mg (MiniMac) on the Upper Arm for 30 Minutes in Healthy Volunteers (Treatment C) (Pharmacokinetic Population)
- Table 14.2.1.8 Plasma Zolmitriptan Pharmacokinetic Parameters for Intranasal Zolmitriptan 2.5 mg in Healthy Volunteers (Treatment D) (Pharmacokinetic Population)
- Table 14.2.1.9 Intervals (Hours) Used for Determination of Plasma
  Zolmitriptan Kel Values for M207 3.8 mg (Sled) on the
  Upper Arm for 30 Minutes in Healthy Volunteers
  (Treatment A) (Pharmacokinetic Population)
- Table 14.2.1.10 Intervals (Hours) Used for Determination of Plasma
  Zolmitriptan Kel Values for M207 3.8 mg (MACAP) on the
  Upper Arm for 30 Minutes in Healthy Volunteers
  (Treatment B) (Pharmacokinetic Population)
- Table 14.2.1.11 Intervals (Hours) Used for Determination of Plasma
  Zolmitriptan Kel Values for M207 3.8 mg (MiniMac) on the
  Upper Arm for 30 Minutes in Healthy Volunteers
  (Treatment C) (Pharmacokinetic Population)
- Table 14.2.1.12 Intervals (Hours) Used for Determination of Plasma
  Zolmitriptan Kel Values for Intranasal Zolmitriptan 2.5 mg in
  Healthy Volunteers (Treatment D) (Pharmacokinetic
  Population)
- Table 14.2.1.13 Relative Bioavailability Between Each Treatment for 3
  Different Formulations of M207 3.8 mg on the Upper Arm
  for 30 Minutes and Intranasal Zolmitriptan 2.5 mg in Healthy
  Volunteers (Pharmacokinetic Population)
- Table 14.2.1.14 Residual Amounts of Zolmitriptan in M207 Patches and on Skin Swabs for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes in Healthy Volunteers (Treatment A) (Pharmacokinetic Population)
- Table 14.2.1.15 Residual Amounts of Zolmitriptan in M207 Patches and on Skin Swabs for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes in Healthy Volunteers (Treatment B) (Pharmacokinetic Population)
- Table 14.2.1.16 Residual Amounts of Zolmitriptan in M207 Patches and on Skin Swabs for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes in Healthy Volunteers (Treatment C) (Pharmacokinetic Population)

## 14.2.2 Plasma Zolmitriptan Figures

- Figure 14.2.2.1 Arithmetic Mean (SD) Plasma Zolmitriptan Concentration
  Versus Time Profiles for 3 Different Formulations of M207
  3.8 mg on the Upper Arm for 30 Minutes and Intranasal
  Zolmitriptan 2.5 mg in Healthy Volunteers (Predose to
  24 Hours Postdose) (Linear Scale) (Pharmacokinetic
  Population)
- Figure 14.2.2.2 Arithmetic Mean (SD) Plasma Zolmitriptan Concentration
  Versus Time Profiles for 3 Different Formulations of M207
  3.8 mg on the Upper Arm for 30 Minutes and Intranasal
  Zolmitriptan 2.5 mg in Healthy Volunteers (Predose to
  2 Hours Postdose) (Linear Scale) (Pharmacokinetic
  Population)
- Figure 14.2.2.3 Arithmetic Mean Plasma Zolmitriptan Concentration Versus
  Time Profiles for 3 Different Formulations of M207 3.8 mg
  on the Upper Arm for 30 Minutes and Intranasal Zolmitriptan
  2.5 mg in Healthy Volunteers (Predose to 24 Hours Postdose)
  (Linear Scale) (Pharmacokinetic Population)
- Figure 14.2.2.4 Mean Plasma Zolmitriptan Concentration Versus Time
  Profiles for 3 Different Formulations of M207 3.8 mg on the
  Upper Arm for 30 Minutes and Intranasal Zolmitriptan
  2.5 mg in Healthy Volunteers (Predose to 2 Hours Postdose)
  (Linear Scale) (Pharmacokinetic Population)

### 14.2.3 Plasma N-Desmethyl Zolmitriptan Tables

- Table 14.2.3.1 Plasma N-Desmethyl Zolmitriptan Concentrations (pg/mL) for M207 3.8 mg (Sled) on the Upper Arm for 30 Minutes in Healthy Volunteers (Treatment A) (Pharmacokinetic Population)
- Table 14.2.3.2 Plasma N-Desmethyl Zolmitriptan Concentrations (pg/mL) for M207 3.8 mg (MACAP) on the Upper Arm for 30 Minutes in Healthy Volunteers (Treatment B) (Pharmacokinetic Population)
- Table 14.2.3.3 Plasma N-Desmethyl Zolmitriptan Concentrations (pg/mL) for M207 3.8 mg (MiniMac) on the Upper Arm for 30 Minutes in Healthy Volunteers (Treatment C) (Pharmacokinetic Population)
- Table 14.2.3.4 Plasma N-Desmethyl Zolmitriptan Concentrations (pg/mL) for Intranasal Zolmitriptan 2.5 mg in Healthy Volunteers (Treatment D) (Pharmacokinetic Population)
- Table 14.2.3.5 Plasma N-Desmethyl Zolmitriptan Pharmacokinetic Parameters for M207 3.8 mg (Sled) on the Upper Arm for

- 30 Minutes in Healthy Volunteers (Treatment A) (Pharmacokinetic Population)
- Table 14.2.3.6 Plasma N-Desmethyl Zolmitriptan Pharmacokinetic Parameters for M207 3.8 mg (MACAP) on the Upper Arm for 30 Minutes in Healthy Volunteers (Treatment B) (Pharmacokinetic Population)
- Table 14.2.3.7 Plasma N-Desmethyl Zolmitriptan Pharmacokinetic
  Parameters for M207 3.8 mg (MiniMac) on the Upper Arm
  for 30 Minutes in Healthy Volunteers (Treatment C)
  (Pharmacokinetic Population)
- Table 14.2.3.8 Plasma N-Desmethyl Zolmitriptan Pharmacokinetic Parameters for Intranasal Zolmitriptan 2.5 mg in Healthy Volunteers (Treatment D) (Pharmacokinetic Population)
- Table 14.2.3.9 Intervals (Hours) Used for Determination of Plasma
  N-Desmethyl Zolmitriptan Kel Values for M207 3.8 mg
  (Sled) on the Upper Arm for 30 Minutes in Healthy
  Volunteers (Treatment A) (Pharmacokinetic Population)
- Table 14.2.3.10 Intervals (Hours) Used for Determination of Plasma
  N-Desmethyl Zolmitriptan Kel Values for M207 3.8 mg
  (MACAP) on the Upper Arm for 30 Minutes in Healthy
  Volunteers (Treatment B) (Pharmacokinetic Population)
- Table 14.2.3.11 Intervals (Hours) Used for Determination of Plasma
  N-Desmethyl Zolmitriptan Kel Values for M207 3.8 mg
  (MiniMac) on the Upper Arm for 30 Minutes in Healthy
  Volunteers (Treatment C) (Pharmacokinetic Population)
- Table 14.2.3.12 Intervals (Hours) Used for Determination of Plasma
  N-Desmethyl Zolmitriptan Kel Values for Intranasal
  Zolmitriptan 2.5 mg in Healthy Volunteers (Treatment D)
  (Pharmacokinetic Population)

## 14.2.4 Plasma N-Desmethyl Zolmitriptan Figures

- Figure 14.2.4.1 Mean (SD) Plasma N-Desmethyl Zolmitriptan Concentration Versus Time Profiles for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes and Intranasal Zolmitriptan 2.5 mg in Healthy Volunteers (Linear Scale) (Pharmacokinetic Population)
- Figure 14.2.4.2 Mean Plasma N-Desmethyl Zolmitriptan Concentration
  Versus Time Profiles for 3 Different Formulations of M207
  3.8 mg on the Upper Arm for 30 Minutes and Intranasal
  Zolmitriptan 2.5 mg in Healthy Volunteers (Linear Scale)
  (Pharmacokinetic Population)

## 14.3 Safety Data Summary Tables and Figures

## 14.3.1 Displays of Adverse Events

- Table 14.3.1.1 Treatment-Emergent Adverse Event Frequency by Treatment
   Number of Subjects Reporting the Event (% of Subject Dosed) (Safety Population)
- Table 14.3.1.2 Treatment-Emergent Adverse Event Frequency by Treatment
   Number of Adverse Events (% of Total Adverse Events)
  (Safety Population)
- Table 14.3.1.3 Treatment-Emergent Adverse Event Frequency by
  Treatment, Severity, and Relationship to Drug Number (%)
  of Subjects Reporting the Event (Safety Population)

## 14.3.2 Listings of Deaths, other Serious and Significant Adverse Events

Table 14.3.2.1 Serious Adverse Events (Safety Population)

# 14.3.3 Narratives of Deaths, other Serious and Certain other Significant Adverse Events

## 14.3.4 Abnormal Laboratory Value Listing (each patient)

- Table 14.3.4.1 Out-of-Range Clinical Laboratory Values and Recheck Results (Safety Population)
- Table 14.3.4.2 Clinically Significant Values According to PI and Recheck Results (Safety Population)

# 14.3.5 Displays of Other Laboratory, Vital Signs, Electrocardiogram, Physical Examination, and Other Safety Data

# 14.3.5.1 Vital Sign, Electrocardiogram and Investigator Visual Skin Assessment Tables

- Table 14.3.5.1.1 Vital Sign Summary and Change From Baseline (Safety Population)
- Table 14.3.5.1.2 12-Lead Electrocardiogram Summary and Change From Baseline (Safety Population)
- Table 14.3.5.1.3 Frequency Counts of Investigator Visual Skin Assessment (Safety Population)
- Table 14.3.5.1.4 Summary of Investigator Visual Skin Assessment (Safety Population)

### 14.3.5.2 Investigator Visual Skin Assessment Figures

- Figure 14.3.5.2.1 Mean Investigator Visual Erythema Assessment Scale by Time Profile (Safety Population)
- Figure 14.3.5.2.2 Mean Investigator Visual Edema Assessment Scale by Time Profile (Safety Population)
- Figure 14.3.5.2.3 Mean Investigator Visual Bruising Assessment Scale by Time Profile (Safety Population)
- Figure 14.3.5.2.4 Mean Investigator Visual Bleeding Assessment Scale by Time Profile (Safety Population)

## 9.3 Section 16 Data Listings

Note: Hepatitis and HIV results that are provided by the clinical laboratory will not be presented in subject data listings and will not be included in any database transfer.

Data listings are numbered following the ICH structure but may be renumbered as appropriate during the compilation of the TFLs for the CSR. The following is a list of appendix numbers and titles that will be included as data listings:

### 16.1 Study Information

Appendix 16.1.9 Statistical Methods

Appendix 16.1.10.1 Clinical Laboratory Reference Ranges

### 16.2 Subject Data Listings

### 16.2.1 Subject Discontinuation

Appendix 16.2.1 Subject Discontinuation (All Randomized Subjects)

#### 16.2.2 Protocol Deviations

Appendix 16.2.2 Protocol Deviations

### 16.2.3 Subjects Excluded from Pharmacokinetic Analysis

Appendix 16.2.3 Subjects Excluded from Pharmacokinetic Analysis

Note: Appendices 16.2.2 and 16.2.3 are generated in MS Word for inclusion in the study report.

### 16.2.4 Demographic Data

| Appendix 16.2.4.1 | Demographics (Safety Population) |
|---|---|
| Appendix 16.2.4.2 | Physical Examination Abnormal Findings (Safety |
| | Population) |
| Appendix 16.2.4.3 | Medical and Surgical History (Safety Population) |
| Appendix 16.2.4.4 | Substance Use (Safety Population) |
| 16.2.5 Compliance | e and/or Drug Concentration Data |
| Appendix 16.2.5.1.1 | Inclusion Criteria |
| Appendix 16.2.5.1.2 | Exclusion Criteria |
| Appendix 16.2.5.2 | Subject Eligibility (Safety Population) |
| Appendix 16.2.5.3 | Check-in Responses (Safety Population) |
| Appendix 16.2.5.4 | Test Compound Administration Times (Safety Population) |
| Appendix 16.2.5.5 | Blood Draw Times (Safety Population) |
| Appendix 16.2.5.6 | Meal Times (Safety Population) |
| Appendix 16.2.5.7 | Prior and Concomitant Medications (Safety Population) |
| 16.2.6 Individual | Pharmacokinetic Response Data |
| Appendix 16.2.6.1 | Plasma Zolmitriptan Concentration Versus Time<br>Profiles for Subject <x> for 3 Different Formulations<br/>of M207 3.8 mg on the Upper Arm for 30 Minutes and<br/>Intranasal Zolmitriptan 2.5 mg (Linear Scale)</x> |
| Appendix 16.2.6.2 | Plasma N-Desmethyl Zolmitriptan Concentration<br>Versus Time Profiles for Subject <x> for 3 Different<br/>Formulations of M207 3.8 mg on the Upper Arm for 30<br/>Minutes and Intranasal Zolmitriptan 2.5 mg (Linear<br/>Scale)</x> |
| Appendix 16.2.6.3 | Residual Amounts of Zolmitriptan in M207 Patches for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes and Intranasal Zolmitriptan 2.5 mg (Safety Population) |
| Appendix 16.2.6.4 | Residual Amounts of Zolmitriptan on Skin Swabs for 3<br>Different Formulations of M207 3.8 mg on the Upper<br>Arm for 30 Minutes and Intranasal Zolmitriptan 2.5 mg<br>(Safety Population) |
| 16.2.7 Adverse Ev | ents Listings |
| Appendix 16.2.7.1.1 | Adverse Events (I of II) (Safety Population) |
| Appendix 16.2.7.1.2 | Adverse Events (II of II) (Safety Population) |
| Appendix 16.2.7.2 | Adverse Event Non-Drug Therapy (Safety Population) |

# 16.2.8 Listings of Individual Laboratory Measurements and Other Safety Observations

| Appendix 16.2.8.1.1 | Clinical Laboratory Report - Serum Chemistry (Safety Population) |
|---|---|
| Appendix 16.2.8.1.2 | Clinical Laboratory Report - Hematology (Safety Population) |
| Appendix 16.2.8.1.3 | Clinical Laboratory Report - Urinalysis (Safety Population) |
| Appendix 16.2.8.1.4 | Clinical Laboratory Report - Urine Drug Screening (Safety Population) |
| Appendix 16.2.8.1.5 | Clinical Laboratory Report - Comments (Safety Population) |
| Appendix 16.2.8.2 | Vital Signs (Safety Population) |
| Appendix 16.2.8.3 | 12-Lead Electrocardiogram (Safety Population) |
| Appendix 16.2.8.4 | Investigator Visual Skin Assessments (Safety Population) |

### 10. TABLE AND FIGURE SHELLS

The following table shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the tables that will be presented and included in the final report. Unless otherwise noted, all in-text tables will be presented in Times New Roman font size 9 and all post-text tables will be presented in Courier New font size 9. These tables will be generated off of the Celerion AdaM Model 2.1 and AdaM Implementation Guide 1.1.

#### **In-text Summary Tables Shells** 10.1

In-text Table 10-1 will be in the following format:

**Subject Disposition Summary Table 10-1** 

| | Rai | | | | |
|---|---|---|---|---|---|
| Disposition | ABDC | BCAD | CDBA | DACB | Overall |
| Enrolled<br>(Randomized) | XX (100%) | XX (100%) | XX (100%) | XX (100%) | XX (100%) |
| Safety Population | XX (100%) | XX (100%) | XX (100%) | XX (100%) | XX (100%) |
| Completed Study | X (X.X%) | X (X.X%) | X (X.X%) | X (X.X%) | X (X.X%) |
| Discontinued Early | X (X,X%) | X (X.X%) | X (X.X%) | X (X.X%) | X (X.X%) |
| <reason1></reason1> | X (X.X%) | X (X.X%) | X (X.X%) | X (X.X%) | X (X.X%) |
| <reason2></reason2> | X (X.X%) | X (X,X%) | X (X.X%) | X (X.X%) | X (X.X%) |

Treatment A: < description>

Treatment B: < description>
Treatment C: < description>
Treatment D: < description>

<AE =Adverse event >

Source: Table 14.1.1

Program: /CAXXXX/sas\_prg/stsas/intexttest/t\_disp.sas\_DDMMMYYYY\_HH:MM

In-text Table 11-1 will be in the following format:

**Table 11-1 Demographic Summary** 

| | | Randomized Treatment Sequence | | | | |
|---|---|---|---|---|---|---|
| Trait | Category/Statistics | ABDC | BCAD | CDBA | DACB | Overall |
| Sex | Male | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Female | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Race | Asian | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | American Indian or<br>Alaska Native | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Black or African<br>American | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Native Hawaiian or<br>Pacific Islander | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | White | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Ethnicity | Hispanic or Latino | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| | Not Hispanic or<br>Latino | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Age* (yrs) | n | XX | XX | XX | XX | XX |
| | Mean | XX.X | XX.X | XX.X | XX.X | XX.X |
| | SD | X.XX | X.XX | X.XX | X.XX | X,XX |
| | Minimum | XX | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX,X | XX.X | XX.X |
| | Maximum | XX | XX | XX | XX | XX |

Treatment A: < description>

Treatment B: < description>
Treatment C: < description>
Treatment D: < description>

BMI = Body mass index

\*Age is derived from birth date to date of informed consent.

Program: /CAXXXXX/sas\_prg/stsas/intexttest/t\_dem.sas DDMMMYYYY HH:MM

Programmer Notes: Height (cm), Weight(kg), and BMI (kg/m²) at screening will be also summarized in the table above.

Table 11-2 Summary of Plasma Zolmitriptan Pharmacokinetics for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes and Intranasal Zolmitriptan 2.5 mg in Healthy Volunteers

| Pharmacokinetic | M207 3.8 mg | M207 3.8 mg | M207 3.8 mg | Zołmitriptan 2.5 mg |
|---|---|---|---|---|
| Parameters | (Sled) | (MACAP) | (MiniMac) | (Intranasal) |
| AUC0-30min (pg•hr/mL) | XXX.X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) |
| | [n=xx] | [n=xx] | [n=xx] | [n=xx] |
| AUC0-60min (pg•hr/mL) | XXX.X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) |
| , | [n=xx] | [n=xx] | [n=xx] | [n=xx] |
| AUC0-120min (pg•hr/mL) | XXX.X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) |
| , | [n=xx] | [n=xx] | [n=xx] | [n=xx] |
| AUC0-t (pg-hr/mL) | XXX.X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) |
| , | [n=xx] | [n=xx] | [n=xx] | [n=xx] |
| AUCO-inf (pg•hr/mL) | XXX.X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) |
| | [n=xx] | [n=xx] | [n≔xx] | [n=xx] |
| Cmax (pg/mL) | XXX.X (XX.X) | XXX.X (XX.X) | XXX,X (XX.X) | XXX.X (XX.X) |
| 4.5 | [n=xx] | [n=xx] | [n=xx] | [n=xx] |
| Tmax (hr) | XXX.X (XX.X, XX.X) | XXX.X (XX.X, XX.X) | XXX.X (XX.X, XX.X) | XXX.X (XX.X, XX.X) |
| , , | [n=xx] | [n=xx] | [n=xx] | [n=xx] |
| t½ (hr) | XXX,X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) |
| ` , | [n=xx] | [n=xx] | [n=xx] | [n=xx] |
| Kel (1/hr) | XXX,X (XX.X) | XXX,X (XX.X) | XXX.X (XX.X) | XXX.X (XX.X) |
| • • | [n=xx] | [n=xx] | [n≕xx] | [n=xx] |

M207 3.8 mg (Sled); M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "Sled" coater and packaged in foil pouches (Treatment A)

M207 3.8 mg (MACAP): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "MACAP" coater and packaged in foil cups (Treatment B)

M207 3.8 mg (MiniMac): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "MiniMac" coater and packaged in foil cups (Treatment C)

Zolmitriptan 2.5 mg (Intranasal): Zolmitriptan 2.5 mg administered intranasally as a single 2.5 mg/0.1 mL spray (Treatment D) AUC and Cmax values are presented as geometric mean and geometric CV%.

Tmax values are presented as median (min, max).

Other parameters are presented as arithmetic mean (± SD).

NA = Not applicable

Source: Tables 14.2.1.5 to 14.2.1.8

#### Notes for Generating the Actual Table:

Presentation of Data:

- n will be presented as an integer (with no decimal). If n is the same for all parameters
  within a given treatment for all 4 treatments, the n will be presented in the treatment
  header only.
- Summary statistics will be presented with same precision as defined in post-text shells

Celerion Note: Per study design needs, the following changes are made to this table relative to Celerion's standard shell: Two additional treatment columns were added.

Program: /CAXXXXX/sas\_prg/pksas/intext-pk-tables.sas DDMMYYYY HH:MM
Program: /CAXXXXX/sas\_prg/pksas/adam\_intext\_pkparam.sas DDMMYYYY HH:MM

Table 11-3 Relative Bioavailability Between Each Treatment for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes and Intranasal Zolmitriptan 2.5 mg in Healthy Volunteers

| Pharmacokinetic Parameters | Geom Mean (Geom CV%) |
|----------------------------|----------------------|
| %Frel(A/B) (%) | XXX.X (XX.X) [n=xx] |
| %Frel(A/C) (%) | XXX.X (XX.X) [n=xx] |
| %Frel(A/D) (%) | XXX.X (XX.X) [n=xx] |
| %Frel(B/C) (%) | XXX.X (XX.X) [n=xx] |
| %Frel(B/D) (%) | XXX.X(XX.X)[n=xx] |
| %Frel(C/D) (%) | XXX.X (XX.X) [n=xx] |

M207 3.8 mg (Sled): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "Sled" coater and packaged in foil pouches (Treatment A)

M207 3.8 mg (MACAP): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "MACAP" coater and packaged in foil cups (Treatment B)

M207 3.8 mg (MiniMac): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "MiniMac" coater and packaged in foil cups (Treatment C)

Zolmitriptan 2.5 mg (Intranasal): Zolmitriptan 2.5 mg administered intranasally as a single 2.5 mg/0.1 mL spray (Treatment D) Source: Table 14.2.1.13

### Notes for Generating the Actual Table:

Presentation of Data:

- n will be presented as an integer (with no decimal). If n is the same for all parameters, the n will be presented along with the "Geom Mean (Geom CV%)" header.
- Geom Mean and Geom CV% will be presented with same precision as defined in post-text shells

Celerion Note: Per study design needs, the following changes are made to this table relative to Celerion's standard shell: One column was deleted.

Program: /CAXXXXX/sas\_prg/pksas/intext-pk-tables.sas DDMMYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/adam\_intext\_pkparam.sas DDMMYYYY HH:MM

Residual Amounts of Zolmitriptan in M207 Patches and on Skin Swabs **Table 11-4** for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes in Healthy Volunteers

| PharmacokineticParameters | M207 3.8 mg (Sled) | M207 3.8 mg (MACAP) | M207 3.8 mg (MiniMac) |
|---|---|---|---|
| Residual Amount in Both Patches Combined (mg) | XX.X(XX.X)[n=xx] | XX.X (XX.X) [n=xx] | XX.X (XX.X) [n=xx] |
| Residual Amount on Both Skin Surfaces Combined (mg) | XX.X (XX.X) [n=xx] | XX.X (XX.X) [n=xx] | XX.X (XX.X) [n=xx] |
| | | XX.X (XX.X) [n=xx] | XX.X (XX.X) [n=xx] |
| M207 3.8 mg (Sled): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "Sled" coater | | | |

and packaged in foil pouches (Treatment A) M207 3.8 mg (MACAP); M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a

"MACAP" coater and packaged in foil cups (Treatment B)

M207 3.8 mg (MiniMac): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "MiniMac" coater and packaged in foil cups (Treatment C)

Actual Dose Administered = Nominal Dose - Residual Amount in Both Patches Combined - Residual Amount on Both Skin Surfaces Combined

Source: Tables 14.2.1.14 to 14.2.1.16

#### Notes for Generating the Actual Table:

#### Presentation of Data:

- n will be presented as an integer (with no decimal). If n is the same for all parameters within a given treatment for all 3 treatments, the n will be presented in the treatment header only.
- Summary statistics will be presented with same precision as defined in post-text shells

Celerion Note: Per study design needs, the following changes are made to this table relative to Celerion's standard shell: One additional treatment column was added.

DDMMYYYYY HH:MM Program: /CAXXXXX/sas prg/pksas/intext-pk-tables.sas Program: /CAXXXXX/sas prg/pksas/adam intext\_pkparam.sas DDMMMYYYY HH:MM In-text Table 12-1 will be in the following format:

Treatment-Emergent Adverse Event Frequency by Treatment - Number **Table 12-1** of Subjects Reporting the Event (% of Subjects Dosed)

| | Treatment | | | | |
|---|---|---|---|---|---|
| Adverse Event* | M207 3.8 mg<br>(Sled) | M207 3.8 mg<br>(MACAP) | M207 3.8 mg<br>(MiniMac) | Zolmitriptan 2.5 mg<br>(Intranasal) | Overall |
| Number of Subjects Dosed | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| Number of Subjects With TEAEs | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) | XX (XX%) |
| System Organ Class 1 | X (X%) | X (X%) | X (X%) | X (X%) | X (X%) |
| Preferred Term 1 | X (X%) | X (X%) | X (X%) | X (X%) | X (X%) |
| Preferred Term 2 | X (X%) | X (X%) | X (X%) | X (X%) | X (X%) |
| System Organ Class 2 | X (X%) | X (X%) | X (X%) | X (X%) | X (X%) |
| Preferred Term I | X (X%) | X (X%) | X (X%) | X (X%) | X (X%) |
| Preferred Term 2 | X (X%) | X (X%) | X (X%) | X (X%) | X (X%) |

M207 3.8 mg (Sled): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "Sled" coater and packaged in foil pouches (Treatment A)
M207 3.8 mg (MACAP): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on

a "MACAP" coater and packaged in foil cups (Treatment B)
M207 3.8 mg (MiniMac): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "MiniMac" coater and packaged in foil cups (Treatment C)

Zolmitriptan 2.5 mg (Intranasal): Zolmitriptan 2.5 mg administered intranasally as a single 2.5 mg/0.1 mL spray (Treatment D) \*Adverse events are coded using MedDRA® Version 20.1.

If a subject has 2 or more clinical adverse events, the subject is counted only once within a category. The same subject may appear in different categories.

TEAEs = Treatment-emergent adverse events

Source: Table 14.3.1.1

Program: /CAXXXXX/sas\_prg/stsas/intexttest/t\_ae.sas DDMMMYYYY HH:MM

## 10.2 Figures Shells

Figures 11-1 to 11-3, 14.2.2.1, 14.2.2.2, and 14.2.4.1 will be in the following format:

Figure 11-1 Arithmetic Mean (SD) Plasma Zolmitriptan Concentration-Time Profiles for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes and Intranasal Zolmitriptan 2.5 mg in Healthy Volunteers (Predose to 24 Hours Postdose)



### Notes:

- Titles of Figures 14.2.2.1, 14.2.2.2, and 14.2.4.1 will include: "(Pharmacokinetic Population)".
- Legend will include: "M207 3.8 mg (Sled)", "M207 3.8 mg (MACAP)", "M207 3.8 mg (MiniMac)", and "Zolmitriptan 2.5 mg (Intranasal)".
- Y-axis labels will be:
  - o Figures 11-1, 11-2, 14.2.2.1, and 14.2.2.2: "Plasma Zolmitriptan Concentration (pg/mL)".
  - o Figures 11-3 and 14.2.4.1: "Plasma N-Desmethyl Zolmitriptan Concentration (pg/mL)".
- Plots for Treatments B, C, and D will be shifted to the right for ease of reading and the following footer will be added: "Plots for Treatments B, C, and D are shifted to the right for ease of reading."

Figures 14.2.2.3, 14.2.2.4, and 14.2.4.2 will be in the following format:

## Figure 14.2.2.3

Arithmetic Mean Plasma Zolmitriptan Concentration Versus Time Profiles for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes and Intranasal Zolmitriptan 2.5 mg in Healthy Volunteers (Predose to 24 Hours Postdose) (Linear Scale) (Pharmacokinetic Population)



Program: /CAXXXXX/sas\_prg/pksas/adam\_meangraph.sas DDMMMYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/meangraph.sas DDMMMYYY HH:MM

#### Notes:

- Legend will include: "M207 3.8 mg (Sled)", "M207 3.8 mg (MACAP)", "M207 3.8 mg (MiniMac)", and "Zolmitriptan 2.5 mg (Intranasal)".
- Y-axis labels will be:
  - o Figures 14.2.2.3 and 14.2.2.4: "Plasma Zolmitriptan Concentration (pg/mL)".
  - o Figure 14.2.4.2: "Plasma N-Desmethyl Zolmitriptan Concentration (pg/mL)".
Figures 12-1 to 12-4 and 14.3.5.2.1 to 14.3.5.2.4 will be in the following format:

Figure 14.3.5.2.1

Mean Investigator Visual Erythema Assessment Scale by Time Profile (Safety Population)



### Notes for Generating the Actual Individual Figure:

- Legend will include: "M207 3.8 mg (Sled)", "M207 3.8 mg (MACAP)", and "M207 3.8 mg (MiniMac)".
- Y-axis label will be:
  - o Figure 12-1 and 14.3.5.2.1: "Investigator Visual Erythema Assessment Scale".
  - o Figure 12-2 and 14.3.5.2.2: "Investigator Visual Edema Assessment Scale".
  - o Figure 12-3 and 14.3.5.2.3: "Investigator Visual Bruising Assessment Scale".
  - o Figure 12-4 and 14.3.5.2.4: "Investigator Visual Bleeding Assessment Scale".

Program: /CAXXXX/sas\_prg/pksas/indgraph-all.sas DDMMYYYY HH:MM
Program: /CAXXXX/sas\_prg/pksas/adam\_indgraph.sas DDMMYYYY HH:MM

Appendices 16.2.6.1 and 16.2.6.2 will be in the following format:

### Appendix 16.2.6.1

Plasma Zolmitriptan Concentration Versus Time Profiles for Subject <X> for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes and Intranasal Zolmitriptan 2.5 mg (Linear Scale)



### Notes for Generating the Actual Individual Figure:

- Legend will include: "M207 3.8 mg (Sled)", "M207 3.8 mg (MACAP)", "M207 3.8 mg (MiniMac)", and "Zolmitriptan 2.5 mg (Intranasal)".
- Y-axis label will be:
  - o Appendix 16.2.6.1: "Plasma Zolmitriptan Concentration (pg/mL)".
  - Appendix 16.2.6.2: "Plasma N-Desmethyl Zolmitriptan Concentration (pg/mL)".

Program: /CAXXXX/sas\_prg/pksas/indgraph-all.sas DDMMYYYY HH:MM
Program: /CAXXXX/sas\_prg/pksas/adam\_indgraph.sas DDMMYYYY HH:MM

### 10.3 Section 14 Summary Tables Shells

Table 14.1.1 will be in the following format:

Table 14.1.1 Summary of Disposition (All Randomized Subjects)

Part 1 of X

Randomized Treatment Sequence

| Category | ABDC | BCAD | CDBA | DACB | Overall |
|---|---|---|---|---|---|
| Enrolled (Randomized)<br>Safety Population<br>Completed Study<br>Discontinued Early<br><reason1></reason1> | XX (100%) XX (100%) X (X%) X (X%) X (X%) X (X%) X (X%) | XX (100%) XX (100%) X (X%) X (X%) X (X%) X (X%) X (X%) | XX (100%) XX (100%) X (X%) X (X%) X (X%) X (X%) X (X%) | XX (100%) XX (100%) X (X%) X (X%) X (X%) X (X%) X (X%) | XX (100%)<br>XX (100%)<br>X (X%)<br>X (X%)<br>X (X%)<br>X (X%)<br>X (X%) |

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >
<AE = Adverse event>

Program: /CAXXXXX/sas\_prg/stsas/tab programname.sas DDMMMYYYY HH:MM

Table 14.1.2 will be in the following format:

Table 14.1.2 Subject Dosing Status and Study Disposition (Safety Population)

Page X of X

| - | Date | DDMMYYYY | DDMMXXXX | DDWWYYYY | DDMMXXXX | DDMMXXXX | DDWWXXXX | | |
|---|---|---|---|---|---|---|---|---|---|
| 440 | study completion<br>Status | Completed Study | Terminated Study Prematurely | Completed Study | Completed Study | Completed Study | Completed Study | | |
| | Q | Yes | Yes | Yes | Yes | Yes | Yes | | × |
| ed | C D | Yes | S<br>N | Yes | Yes | Yes | Yes | - | × |
| Dosed | Э | Yes | Yes | Yes | Yes | Yes | Yes | | × |
| | A. | Yes | Yes | Yes | Yes | Yes | Yes | | × |
| E | realment<br>Sequence | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | | |
| -<br>-<br>- | Number | <br> <br> <br> <br> | × | × | × | × | × | | |

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >

Program: /CPXXXXX/sas\_prg/stsas/tab\_PROGRAMMPME.sas DDMMMYYYY HH:MM

Table 14.1.3 will be in the following format:

Table 14.1.3 Demographic Summary (Safety Population)

×

Page 1 of

| Sequence |
|------------|
| Treatment |
| Randomized |

| Trait | | ABDC | BC | BCAD | C | CDBA | ă | DACB | 0 | Overall |
|---|---|---|---|---|---|---|---|---|---|---|
| Sex | Male | X (XX%) | ) × | (XX%) | × | X (XX%) | į × | X (XX%) | × | X (XX8) |
| | Female | X (XX%) | × | (XX%) | × | (XX%) | × | (XX%) | × | (XX%) |
| Race | American Indian or | X (XX%) | × | (XX%) | × | ( XX % ) | × | ( %XX ) X | × | (XX%) |
| | Alaska native<br>Asian | X (XX%) | | XX%) | | XX%) | | (XX%) | × | (XX%) |
| | Black or African American | X (XX%) | | (XX%) | × | (XX%) | × | (XX%) | × | (XX%) |
| | Native Hawaiian or<br>Pacific Islander | X (XX%) | × | (XX%) | × | (XX%) | × | (XX%) | × | (XX%) |
| | White | X (XX%) | × | (XX%) | × | (XX%) | × | X (XX%) | × | (XX%) |
| Ethnicity | Hispanic or Latino | X (XX%) | × | XX%) | × | XX%) | × | (XX%) | × | (XX%) |
| | Not Hispanic or Latino | X (XX%) | × | (XX%) | × | (XX%) | × | (XX%) | × | (XX%) |
| Age* (yr) | ជ | × | | × | | × | | × | | × |
| | Mean | ×× | | ×.× | | X.X | | X.X | | × |
| | SD | XX.XX | × | XX | × | XX. | ~ | XX. X | × | XX |
| | Minimum | XX | | XX | | XX | | X | | X |
| | Median | ×× | | X.X | | × | | X.X | | ×.× |
| | Maximum | XX | | XX | | X | | X | | × |

Programmer Note: Height (cm), Weight(kg), and BMI (kg/m²) at screening will be also summarized in the table above. Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMME.sas DDMAMYYY HH:MM

Tables 14.2.1.1 to 14.2.1.4 and 14.2.3.1 to 14.2.3.4 will be in the following format:

Page X of X Table 14.2.1.1. Plasma Zolmitriptan Concentrations (qunits>) for M207 3.8 mg (Sled) on the Upper Arm for 30 Minutes in Healthy Volunteers (Treatment A) (Pharmacokinetic Population)

| Subject | Treatment | Study | | | | Sample | le Times | (Juz.) | | | ' |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Number | Sequence | Period | Predose | × | × | × | × | × | × | × | × |
| X | XXXX | × | BIQ | × | × | × | × | × | × | × | × |
| × | XXXX | × | BIQ | × | × | × | × | × | × | × | × |
| × | XXXX | × | BIQ | × | × | × | × | × | × | × | ¤ |
| Ü. | | | × | × | × | × | × | × | × | × | × |
| Mean | | | XX.X | XX.X | XX.XX | XX.X | XX.X | XX.X | x.x | x.xx | x.xx |
| SD | | | ××.×× | ×.× | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX | XX.XX |
| CV% | | | | ×.× | X.X | ×.× | XX.X | XX.X | ×.× | X.XX | x.xx |
| SEM | | | XX.XX | XX.XX | XX.XX | XX.XX | ×××× | XX.XX | XX.XX | XX.XX | XX.XX |
| Minimum | | | × | × | X | × | × | × | × | × | × |
| Median | | | ×.× | XX.X | X.XX | XX.X | XX.X | XXX | XX | ××× | XX |
| Maximum | | | × | × | × | × | × | × | × | × | × |

N207 3.8 mg (Sled): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "Sled" coater and packaged in foil pouches (Treatment A)

For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of <XX> are treated as <0> before the first quantifiable concentration and as missing elsewhere.

. = Value missing or not reportable.

## Notes for Generating the Actual Table:

Presentation of Data:

Concentrations will be presented to same precision as in bio data.

Summary statistics presentation with respect to the precision of the bio data: n = integer; Mean and Median +1; SD and SEM +2, Min and Max +0, CV% to 1 decimal

Programmer Note:

PK Time points are: Predose and 0.0333, 0.0833, 0.1667, 0.25, 0.3333, 0.5, 0.75, 1, 1.5, 2, 4, 8, 12, and 24 hours postdose. DOMMYYYYY HH: MM

Program: /GAXXXX/sas\_prg/pksas/pk-conc-tables.sas Program: /GAXXXXX/sas\_prg/pksas/pk-conc-tables-sig.sas

/CAXXXX/sas\_prg/pksas/adam\_conc.sas

MYXYYWWWICC

# Tables 14.2.1.5 to 14.2.1.8 and 14.2.3.5 to 14.2.3.8 will be in the following format:

Table 14.2.1.5. Plasma Zolmitriptan Pharmacokinetic Parameters for MZ07 3.8 mg (Sled) on the Upper Arm for 30 Minutes in Healthy Volunteers Page X of X (Treatment A) (Pharmacokinetic Population)

| ( + : m., | x.xx<br>x.xx<br>x.xx<br>x.xx | 7.2 | Period (units) (units) |
|---|---|---|---|
| ∄ | × × × × | | XX.XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX<br>XX.XX |
| | X | | X.XX<br>XXX<br>XXXX<br>XXXX<br>XXXX<br>XXXX |
| | ×× | | XXX<br>XXXX<br>XXXX<br>XXXX<br>XXXX<br>XXXX |
| | ××× | | X.XX<br>XXXX<br>XXXX<br>XXXX<br>XXXX |
| | **** | | X.XX<br>XXX<br>XXX<br>XXX<br>XXX |
| | XX.XX | | XXXX<br>XXX<br>XXXXX |
| | XX.X | | XXX XX |
| | X.X | | |
| | × | | |
| X.XX.X | X.XXX | , | |
| × | XX.XX | , , | , , |
| | XX.X | | |
| × | XX | - | - |
| | × | | |
| × | X.XX | , | , |
| | XX.XX | | |
| × | X.XXX | | |
| | XX | | |

M207 3.8 mg (Sled): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "Sled" coater and packaged in foil pouches (Treatment A)

- Value missing or not reportable.

### Notes for Generating the Actual Table:

### Presentation of Data:

PK Parameters will be presented in the following order and with following units: AUCO-30min (pg\*hr/mL), AUCO-60min (pg\*hr/mL), AUCO-120min (pg\*hr/mL),

### Zosano Pharma Corporation M207, CP-2019-002

## Celerion, Clinical Study Report No. CA27752

- For Tables 14.2.3.5 to 14.2.3.8, AUCO-inf(m/p) will be presented after AUCO-inf.
  - n will be presented as an integer (with no decimal);
- AUCS, CMax, and Kel will be presented with, at maximum, the precision of the bio data, and, at minimum, 3 significant figures (to be determined by the PKist once bio data are received).
- Thax and t1/2 will be presented with 2 decimals. Summary statistics for time-based parameters will be presented as: Mean, Median, and Geom Mean +1; SD +2, Min and Max +0.
- Summary statistics for exposure parameters will be presented as: Mean, Median, and Geom Mean +1; SD and SEM +2, Min and Max +0; CV% and Geom CV% to 1 decimal place.

Program: /CAXXXX/sas\_prg/pksas/pk-tables.sas Program: /CAXXXX/sas\_prg/pksas/adam\_pkparam.sas

DDWMYYYY HH:MM DDWMWYYYY HH:MM

# Tables 14.2.1.9 to 14.2.1.12 and 14.2.3.9 to 14.2.3.12 will be in the following format:

Table 14.2.1.9. Intervals (Hours) Used for Determination of Plasma Zolmitriptan Kel Values for M207 3.8 mg (Sled) on the Upper Arm for 30 Minutes in Healthy Volunteers (Treatment A) (Pharmacokinetic Population) Page X of X

| ជ | × | × | × | × | × | × |
|---|---|---|---|---|---|---|
| <b>%</b> | XXX.X | XXX X | XXXXX | X.XXX | X.XXX | X.XXX |
| Interval | x.x xx.x | XX.X - XX.X | X.X - X.X | XX.X - XX.X | XX.X - XX.X | XX.X - XX.X |
| Treatment | × | × | × | × | × | × |
| Subject<br>Number | × | × | × | × | × | × |

M207 3.8 mg (Sled) = M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "Sled" coater and packaged in foil pouches (Treatment A)  $R^2=$  Coefficient of determination

 $n=\mbox{Number}$  of points used in Kel calculation . = Kel value not reportable.

### Notes for Generating the Actual Table:

Presentation of Data:

Interval start and stop times will be presented to 1 decimal or 3 sig figures min;

R<sup>2</sup> will be presented to 3 decimals;

 $\boldsymbol{n}$  will be presented as an integer (with no decimal).

DDMMYYYYY HH:MM DDMMYYYY HH:MM Program: /CAXXXXX/sas\_prg/pksas/kel-tables-parallel.sas Program: /CAXXXXX/sas\_prg/pksas/adam\_kel.sas DDM

Page X of X Table 14.2.1.13. Relative Bioavailability Between Each Treatment for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes and Intranasal Zolmitriptan 2.5 mg in Healthy Volunteers (Pharmacokinetic Population)

| | param6<br>(units) | XXXX | XXX.X | X.XXX | XXX.X | XXXX | XXXX | X.XXX | × | X.XXXX | XX.XX | XX.X | XX.XX | XXX.X | X.XXXX | X.XXX | X.XXXX | x.x. |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | param5<br>(units) | XX.X | X.X | x.x | x.x | XX.X | ×.× | x.x | XX | XX.XX | XX.XX | XX.X | XX.XX | XX.X | XX.XX | x.x | XX.XX | xx.x |
| eters | param4<br>(units) | XXX | XXX | XXX | XXX | XXX | XX | XXX | × | XXXX.X | XX.XX | ×.× | XX.XX | XXX | XXX.X | XX | x.xx.x | x.xx |
| | param3<br>(units) | XXX | XXX | XXX | XXX | XX | XXX | XXX | XX | xxxx.x | XX.XX | XX.X | XX.XX | XXX | XXX.X | XXX | XXXX.X | XX.X |
| | param2<br>(units) | X.XX | XX.XX | XX.X | XX.X | X.XX | X.XX | x.x | × | XXXXX | XX.XX | xx.x | XX.XX | X.XX | X.XXX | X.XX | X.XXX | xx.x |
| | paraml<br>(units) | XXX | x.x | XXX | X.X | x.x | X.XX | XX | × | XXXX.X | XX.XX | X.XX | XX.XX | X.X | XX.XX | XXX | XXX.X | X.XX |
| | Subject<br>Number | × | × | × | × | × | × | × | ц | Mean | GS . | CV% | SEM | Miniman | Median | Maximum | Geom Mean | Geom CV% |

coater and packaged in foil pouches (Treatment A)
M207 3.8 mg (MACAP): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "MACAP" coater and packaged in foil cups (Treatment B)
M207 3.8 mg (MiniMac): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "WiniMac" coater and packaged in foil cups (Treatment C)
WiniMac" coater and packaged in foil cups (Treatment C)
Zolmitriptan 2.5 mg (Intranasal): Zolmitriptan 2.5 mg administered intranasally as a single 2.5 mg/0.1 mL spray (Treatment D) M207 3.8 mg (Sled): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "Sled" . = Value missing or not reportable.

### Notes for Generating the Actual Table:

### Presentation of Data:

- PK Parameters will be presented in the following order and with following units: %frel(A/B) (%), %Frel(A/C) (%), and %Frel(A/D) (%), and %Frel(C/D) (%).
  - n will be presented as an integer (with no decimal);
    - Parameters will be presented to 1 decimal place.
- Summary statistics for exposure parameters will be presented as: Mean, Median, and Geom Mean +1; SD and SEM +2, Min and Max +0; CV% and Geom CV% to 1 decimal place.

Program: /CAXXXX/sas\_prg/pksas/pk-tables.sas DDMMYYYY HH:NM Program: /CAXXXXX/sas\_prg/pksas/adam\_pkparam.sas DDMMYYYY HH:NM

# Tables 14.2.1.14 to 14.2.1.16 will be in the following format:

Page X of X Table 14.2.1.14. Residual Amounts of Zolmitriptan in MZO7 Patches and on Skin Swabs for 3 Different Formulations of MZO7 3.8 mg on the Upper Arm for 30 Minutes in Healthy Volunteers (Treatment A) (Safety Population)

| Actual Dose Administered (mg) | ×× | XX | XX | X.X | XX.XX | X.X | XX.XX | × | x.xx | × |
|---|---|---|---|---|---|---|---|---|---|---|
| Residual Amount on Skin Swabs (mg) | ×× | 1 × | XX | XX.X | XX.XX | X.X. | XX.XX | XX | XX.X | × |
| Residual Amount in Patches (mg) | × | ¶ X | XX | X.XX | XX.XX | X.XX | XX.XX | × | X.X | X |
| Study<br>Period | ×× | < × | | | | | | | | |
| Treatment<br>Sequence | XXXXX | XXX | | | | | | | | |
| Subject<br>Number | ×× | < ⋈ | ជ | Mean | S | 600 | SEM | Minimim | Median | Maximum |

M207 3.8 mg (Sled): M207 3.8 mg achinistered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "Sled" coater and packaged Residual Amount in patches = Residual armount in both patches combined in foil pouches (Treatment A)

Residual Amount on skin swabs = Residual anmount on both skin surfaces combined

Actual Dose Administered = Nominal Dose - Residual Amount in Patches - Residual Amount on Skin Swabs
For the calculation of summary statistics, values that are below the limit of quantitation (BLQ) of <XX> are treated as <0>.

. = Value missing or not reportable.

### Notes for Generating the Actual Table:

Presentation of Data:

Residual amounts will be presented to same precision as in bio data.

Summary statistics presentation with respect to the precision of the bio data: n = integer; Mean and Median +1; SD and SEM +2, Min and Max +0, CV% to 1 decimal

/CAXXXX/sas\_prg/pksas/adam\_pkparam.sas /CAXXXXX/sas\_prg/pksas/pk-tables.sas Program: Program:

HH:MM 田:風 DDMMMXXXX DDMMMXXXX

Table 14.3.1.1 will be in the following format:

Page 1 of X Table 14.3.1.1 Treatment-Emergent Adverse Event Frequency by Treatment - Number of Subjects Reporting the Event (% of Subjects Dosed) (Safety Population)

Treatment

| Adverse Event* | M207 3.8 mg<br>(Sled) | M207 3.8 mg<br>(MACAP) | Minimac) | Zolmitriptan 2.5 mg<br>(Intranasal) | Overall |
|---|---|---|---|---|---|
| Number of Subjects Dosed<br>Number of Subjects With TEAEs | XX (XXX%)<br>X ( X%) | XX (XXX%)<br>X ( XX%) | XX (XXX%)<br>X (XXX%) | XX (XXX%)<br>X ( XX%) | XX (XXXX%)<br>X (XXXX%) |
| | ( X ) X | X ( X%) | X ( X%) | X ( X%) | X ( X%) |
| Vision blurred | X (X8) | _ | X (X%) | X ( X%) | _ |
| Gastrointestinal disorders | X (X%) | X (X8) | X (X%) | X ( X%) | X ( X%) |
| Dyspepsia | X (X%) | ~ | X ( X%) | X ( X%) | _ |
| Nausea | _ | X (X%) | ~ | _ | _ |
| Musculoskeletal and connective | X (X%) | X (X8) | ~_ | _ | |
| tissue disorders | | | | | |
| Back pain | X (X8) | X (X8) | X (X%) | X ( X%) | X (X%) |
| Muscle cramps | X (X%) | ( | X ( X%) | X ( X%) | X (X8) |
| Musculoskeletal pain | ( 8X ) X | X (X%) | × (×%) | X ( X%) | ( %X ) X |

- made on a - made on patches 30 min wear time (upper arm application)  $\rm M207~3.8~mg$  (Sled): M207 3.8 mg administered as two 1.9 mg "Sled" coater and packaged in foil pouches (Treatment A)

M207 3.8 mg (MACAP): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) a "MACAP" coater and packaged in foil cups (Treatment B)

- made M207 3.8 mg (MiniMac): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) on a "MiniMac" coater and packaged in foil cups (Treatment C)

Zolmitriptan 2.5 mg (Intranasal): Zolmitriptan 2.5 mg administered intranasally as a single 2.5 mg/0.1 mL spray \* Adverse events are coded using MedDRA Version 20.1. (Treatment D)

If a subject has 2 or more clinical adverse events, the subject is counted only once within a category. The same subject may appear in different categories. TEAEs = Treatment-emergent adverse events

Program: /CAXXXXX/sas\_prg/stsas/tab programname.sas DDMMMYYYY HH:NM

Table 14.3.1.2 will be in the following format:


Table 14.3.1.2 Treatment-Emergent Adverse Event Frequency by Treatment - Number of Adverse Events (% of Total Adverse Events) (Safety Population)

Treatment

| Adverse Event* | M207 3.8 mg<br>(Sled) | M207 3.8 mg<br>(MACAP) | 1 | Zolmitriptan 2.5 mg<br>(Intranasal) | Overall |
|---|---|---|---|---|---|
| Number of TEAEs | XX (100%) | XX (100%) | XX (1008) | XX (100%) | XX (100%) |
| Eve disorders | X ( X%) | X (X%) | X ( X%) | į. | X ( X%) |
| Vision blurred | | X (X8) | X ( X%) | | X (X%) |
| Gastrointestinal disorders | X (X%) | X (X%) | X ( X%) | | ( X X ) X |
| Dyspepsia | | X ( X%) | X ( X%) | | X (X%) |
| Nausea | | ( X%) X | X ( X%) | | X (X%) |
| Musculoskeletal and connective | X (X%) | X ( X%) | X ( X%) | X ( X%) | X (X8) |
| tissue disorders | | | | | |
| Back pain | X (X8) | X (X%) | X ( X%) | ( X%) X | X (X8) |
| Muscle cramps | ( X% ) X | X ( X%) | X (X%) | | X (X8) |
| Musculoskeletal pain | ( X X X | ( X%)<br>X | X ( X%) | | ( X%) X |

- made on a made on M207 3.8 mg (Sled): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) "Sled" coater and packaged in foil pouches (Treatment A)
M207 3.8 mg (MACAP): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application)
a "MACAP" coater and packaged in foil cups (Treatment B)

- made M207 3.8 mg (MiniMac): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) on a "MiniMac" coater and packaged in foil cups (Treatment C)
Zolmitriptan 2.5 mg (Intranasal): Zolmitriptan 2.5 mg administered intranasally as a single 2.5 mg/0.1 mL spray

(Treatment D)

DDMMMXXXX /CAXXXXX/sas\_prg/stsas/tab programname.sas Program:

<sup>\*</sup> Adverse events are coded using MedDRA Version 20.1. TEAEs = Treatment-emergent adverse events

Table 14.3.1.3 will be in the following format:

Page 1 of X Table 14.3.1.3 Treatment-Emergent Adverse Event Frequency by Treatment, Severity, and Relationship to Study Drug - Number (%) of Subjects Reporting the Event (Safety Population)

| rent* Treatment TEAES Mild Moderate Severe pain A X X X X X X X X X X X X X X X X X X | | | Number of<br>Subjects | | Severity Grade | Φ | Relations | Relationship to Study Drug | Drug |
|---|---|---|---|---|---|---|---|---|---|
| tion the pain the back of the | Adverse Event* | Treatment | TEAES | Mild | Moderate | Severe | Probably<br>Related | Possibly<br>Related | Not<br>Related |
| ton the back of th | Abdominal pain | #<br> | | i<br> <br> <br> ×<br> | <br> | ;<br>!<br>! × | ι<br> | | <br> |
| thoea C X X X X X X X X X X X X X X X X X X | Constipation | മ | × | × | × | × | × | × | × |
| hoea C X X X X X X X X X X X X X X X X X X | Dry throat | щ | × | × | × | × | × | × | × |
| Jestion B X X X X X X X X X X X X X X X X X X | Oysmenorrhoea | υ | × | × | × | × | × | × | × |
| Jestion B X X X X X X X X X X X X X X X X X X | Dyspepsia | Д | × | × | × | × | × | × | × |
| Jestion B X X X X X X X X X X X X X X X X X X | Headache | υ | × | × | × | × | × | × | × |
| Jestion B X X X X X X X X X X X X X X X X X X | | Д | × | × | × | × | × | × | × |
| Jestion B X X X X X X X X X X X X X X X X X X | Myalgia | ď | × | × | × | × | × | × | × |
| # K | al congestion | д | × | × | × | × | × | × | × |
| # X X X X X X X X X X X X X X X X X X X | Skin laceration | υ | × | × | × | × | × | × | × |
| B | Treatment A | | | :<br>:<br>: × | <br> | i<br> <br> | <br> | ;<br>! | × |
| C | Treatment B | | × | × | × | × | × | × | × |
| D X X X X X X X X X X X X X X X X X X X | Treatment C | | × | × | × | × | × | × | × |
| 1 . x x x x x x x x | Treatment D | | × | × | × | × | × | × | × |
| | Overall | | × | × | × | × | × | × | × |

Treatment A: < > Treatment B:

Treatment C: < >

Treatment D: < >

\* Adverse events are coded using MedDRA Version 20.1. TEAEs = Treatment-emergent adverse events

When a subject experienced the same AE at more than one level of severity during a treatment period, the AE with the maximum severity was counted. When a subject experienced the same AE at more than one level of drug relationship during a treatment period, the most related AE

Program: /CAXXXXX/sas\_prg/stsas/tab programname.sas DDWMMYYYY HH:MM

Table 14.3.2.1 will be in the following format:

Table 14.3.2.1 Serious Adverse Events (Safety Population)

Programmer Note: Will match 16.2.7 or contain the following statement: "There were no serious adverse events recorded chring the study."

Statistical Analysis Plan, 04 July 2019

Program: /CAXXXXX/sas\_prg/stsas/tab\_PROGRAMNAME.sas DIMMATYYY HH:NM

Table 14.3.4.1 Out-of-Range Clinical Laboratory Values and Recheck Results (Safety Population)


| Unit | mg/dL<br>mg/dL<br>mg/dL<br>mg/dL |
|---|---|
| Reference Range | ××××<br> |
| Result | XXX<br>XXX HYR+<br>XXX HY+<br>XXX BN |
| Test | Cholesterol<br>Cholesterol<br>Cholesterol<br>Cholesterol |
| Department | Serum Chemistry<br>Serum Chemistry<br>Serum Chemistry<br>Serum Chemistry |
| Time | HH:MM:SS<br>HH:MM:SS<br>HH:MM:SS<br>HH:MM:SS |
| r Date | XXXXMMMQQ<br>XXXXXMMQQ<br>XXXXXXXX<br>XXXXMMQQ |
| / Hour I | XXXX |
| Day | ×××× |
| ubject Age#/ Study<br>unber Sex Period | × |
| Age#/<br>Sex | X/XX |
| Subject<br>Number | × |

# Age is derived from birth date to date of informed consent. F = Female, M = Male

H = Above reference range, L = Below reference range

Computer: N = Not clinically significant, Y = Clinically significant

PI Interpretation: - = Not clinically significant, R = Recheck requested, ^ = Will be retested later, + = Clinically significant

Replace Parameter1, 2 etc. with actual lab tests in the study. Sort unscheduled assessment and early termination records chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for. Add fourth flag in the cases that ^ or R are used for the PI flag. This flag will be found in the ClinQuick Extraction. Programmer Notes:

Program: /CAXXXXX/sas\_prg/stsas/tab\_FRCGRAMAME.sas DIMMAYYYY HH:NM

Table 14.3.4.2 Clinically Significant Values According to PI and Recheck Results (Safety Population)

| Unit | mg/dī<br>mg/dī<br>mg/dī<br>mg/dī |
|---|---|
| Reference Range | × |
| Result | X HYR+<br>X HY+<br>X HY+<br>X HN |
| Ř | XXXX |
| Test | Cholesterol<br>Cholesterol<br>Cholesterol<br>Cholesterol |
| at a | Serum Chemistry<br>Serum Chemistry<br>Serum Chemistry<br>Serum Chemistry |
| Time Dep | HH:MM:SS<br>HH:MM:SS<br>HH:MM:SS<br>HH:MM:SS |
| Date | ***** |
| Day | ×××× |
| | × |
| Age#/<br>Sex | x/xx |
| Subject Age#/Stu<br>Number Sex Per | × |

# Age is derived from birth date to date of informed consent. F = Female, M = Male

H = Above reference range Computer: Y = Clinically significant

PI Interpretation: R = Recheck requested, + = Clinically significant

Programmer Note: All time points for a subject/test with at least one value deemed as CS by the PI will be presented in this table.

If there were no CS values as deemed by PI (i.e., no "CS" or "Clinically Significant" in the PI flag [3<sup>rd</sup> or 4<sup>th</sup> field] in the laboratory dataset), then this table will contain only the statement: "There were no laboratory values deemed clinically significant by the PI in the study."

/CAXXXXX/sas prg/stsas/tab PRXRAMMPME.sas DDMMNYYY HH:MM

Table 14.3.5.1.1 will be in the following format:

| (Safety Population) |
|---------------------|
| From Baseline |
| Froi |
| Change |
| and |
| Sign Summary |
| Sign |
| Vital |
| <b>:</b> |
| 14.3.5.1 |
| Table |


| Le + 517 | | | | | | Treatment | | | Change | e From Baseline* | seline* |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Sign (unit) | Point | Statistic | Overall | M207<br>3.8 mg<br>(Sled) | M207<br>3.8 mg<br>(MACAP) | M207<br>3.8 mg<br>(MiniMac) | Zolmitrip-<br>tan 2.5 mg<br>(Intranasal) | M207<br>3.8 mg<br>(Sled) | M207<br>3.8 mg<br>(MACAP) | M207 M207<br>3.8 mg 3.8 mg<br>(MACAP) (Minimac) | Zolmitrip-<br>tan 2.5 mg<br>(Intranasal) |
| Testname<br>(unit) | Screening | T I | <br> | <br> | | | | | | # t | |
| \\ \frac{1}{2} \\ \fr | | Mean | х.х | | | | | | | - | |
| | | SD<br>Minimum | ×.<br>×. | | | | | | | | |
| | | Median | X.X | | | | | | | | |
| | | Maximum | X | | | | | | | | |
| | Dav -1 | £ | * | | | | | | | | |
| | 1<br>1 | Mean | : ×: | | | | | | | | |
| | | SD | ×.× | | | | | | | | |
| | | Minimum | X.XX | | | | | | | | |
| | | Maximum | × × × | | | | | | | | |
| | Day 1, | ជ | | | | × | * | | | | |
| | Predose | Mean | | x.x | ×× | ×× | ××× | | | | |
| | | SD | | | | X.XX | X.XX | | | | |
| | | Minimum | | | | X | XX | | | | |
| | | Median | | ××× | ×.× | ×.× | ×.× | | | | |
| | | Maximum | | XX | XX | ×× | XX | | | | |
| | Day 1, | q | | × | × | × | × | × | × | × | × |
| | 10 Min | Mean | | ×.× | ××× | ×.× | X.X | x.x | ×.× | ×× | ×× |
| | | SD | | XX.XX | X.XX | X.XX | X.XX | X.XX | XX.XX | XX.XX | X.XX |
| | | Minimum | | X | XX | XX | XX | × | XX | XX | XX |
| | | Median | | ××× | ×.× | x.x | x.x | ××× | ×.× | x.x | ×.× |
| | | Maximum | | X | XX | XX | XX | X | X | XX | XX |

"Sled" coater and packaged in foil pouches (Treatment A) M207 3.8 mg (MACAP): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on M207 3.8 mg (Sled): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on M207 3.8 mg (MiniMac): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "MiniMac" coater and packaged in foil cups (Treatment C) Zolmitriptan 2.5 mg (Intranasal): Zolmitriptan 2.5 mg administered intranasally as a single 2.5 mg/0.1 mL spray \*Baseline is the last non-missing assessment prior to dosing in each period (Day 1 Predose). Supine and sitting measurement were pooled in the summaries. a "MACAP" coater and packaged in foil cups (Treatment B) (Treatment D)

Programmer Notes: Similar for all time points and vital signs. Change from baseline will not be calculated for the End of Study (Day 3 of Period 4) time point. The End of Study time point will be summarized in the Overall column.

Program: /CAXXXXX/sas\_prg/stsas/tab programname.sas DDMMMYYYY HH:NM

Table 14.3.5.1.2 will be in the following format:

Page 1 of X Table 14.3.5.1.2 12-Lead Electrocardiogram Summary and Change From Baseline (Safety Population)

| 4<br>4<br>4<br>8<br>6 | (<br>E | | | | | Treatment | | | Change | Change From Baseline* | seline* |
|---|---|---|---|---|---|---|---|---|---|---|---|
| (unit) | Point | Statistic | Overall | M207<br>3.8 mg<br>(Sled) | M207<br>3.8 mg<br>(MACAP) | M207<br>3.8 mg<br>(MiniMac) | Zolmitrip-<br>tan 2.5 mg<br>(Intranasal) | M207<br>3.8 mg<br>(Sled) | M207<br>3.8 mg<br>(MACAE) ( | M207<br>3.8 mg<br>MiniMac) | Zolmitrip-<br>tan 2.5 mg<br>(Intranasal) |
| Parameter (unit) | Screening | u | <br> -<br> -<br> -<br> -<br> -<br> -<br> - | | <br> | | · = | | | 1<br>1<br>1<br>1<br>1<br>1<br>1 | |
| | | Mean | ×.× | | | | | | | | |
| | | SD | x.xx | | | | | | | | |
| | | Minimum | X | | | | | | | | |
| | | Median | × | | | | | | | | |
| | i | Maximum | X | | | | | | | | |
| | Day 1, | ជ | | × | × | × | × | | | | |
| | Predose | Mean | | ×.× | ×.× | х.х | X.X | | | | |
| | | SD | | XX.X | X.XX | X.XX | X.XX | | | | |
| | | Minimum | | X | XX | XX | XX | | | | |
| | | Median | | ×.× | ×.× | x.x | ××× | | | | |
| | | Maximum | | XX | XX | × | XX | | | | |
| | Day 1, | ជ | | × | × | × | × | × | × | × | × |
| | 15 Min | Mean | | ×× | ×.× | ×× | х.х | ×.× | ×:× | ×× | ×× |
| | | SD | | XX.X | X.XX | XX.XX | X.XX | XX.XX | xx.x | X.XX | XX.X |
| | | Minimum | | XX | XX | × | XX | ×× | ×× | × | XX |
| | | Median | | ×.× | ×.× | x.x | x.x | ×.× | × | x.x | X.X |
| | | Maximum | | XX | XX | × | XX | X | X | XX | X |

M207 3.8 mg (Sled): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "Sled" coater and packaged in foil pouches (Treatment A)
M207 3.8 mg (MACAP): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "MACAP" coater and packaged in foil cups (Treatment B)
M207 3.8 mg (MiniMac): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "MiniMac" coater and packaged in foil cups (Treatment C)

Zolmitriptan 2.5 mg (Intranasal): Zolmitriptan 2.5 mg administered intranasally as a single 2.5 mg/0.1 mL spray (Treatment D)

\*Baseline is the last non-missing assessment prior to dosing in each period (Day 1 Predose).

Programmer Notes: Similar for all time points and ECG parameters. Change from baseline will not be calculated for the End of Study (Day 3 of Period 4) time point. The End of Study time point will be summarized in the Overall column.

Program: /CAXXXXX/sas\_prg/stsas/tab programname.sas DDMMMYYYY HH:MM

# Table 14.3.5.1.3 will be in the following format:

Table 14.3.5.1.3 Summary of Investigator Visual Skin Assessment (Safety Population)

| , | | | | | | S | Skin Asse | SSm | Assessment Scales* | *<br>() | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Assessment | Treatment | Time Point | Z | <br> <br> | 0 | ļ | 1 | | 2 | | т |
| Erythema | × | Day 1, Predose<br>Day 1, 30 Min<br>Day 1, 60 Min<br>Day 1, 8 Hours<br>Day 2, 24 Hours | *** | ××××× | X (XX.X%)<br>X (XX.X%)<br>X (XX.X%)<br>X (XX.X%)<br>X (XX.X%) | ××××× | X (XX.X%)<br>X (XX.X%)<br>X (XX.X%)<br>X (XX.X%)<br>X (XX.X%) | ××××× | (X.XX%)<br>(X.XX%)<br>(X.XX%)<br>(X.XX%)<br>(X.XX%) | XXXXX | (XX.X%)<br>(XX.X%)<br>(XX.X%)<br>(XX.X%) |

<Similar for all skin assessments, treatments and time points>

Treatment B: < >
Treatment C: < >
Treatment D: < >

N = Number of non-missing observations. Percentages are based on the number of non-missing observations.

At each treatment and time point, the worst assessment scale between the two dosing patches application sites was used in the summaries.

\* Scale descriptions:

Exythems: 0 = Mone; 1 = Mild redness; 2 = Moderate colored redness; 3 = Beet colored redness

Edema: 0 = None; 1 = Slight edema; 2 = Moderate edema; 3 = Severe edema

Bruising (visual rating): 0 = None; 1 = ≤ 25% application site has bruising spots; 2 = ≥ 26 to ≤ 50% application site has bruising spots

3 = > 50% application site has bruising spots

Bleeding: 0 = None; 1 = Pink color on skin; 2 = Visible blood drop; 3 = Active bleeding

Program: /CAXXXXX/sas\_prg/stsas/tab programname.sas DDMMMYYYY HH:NM

Table 14.3.5.1.4 will be in the following format:

Table 14.3.5.1.4 Summary of Investigator Visual Skin Assessment (Safety Population)

×

Page 1 of

| 27.5 | e<br>E | | | Treatment | ıt |
|---|---|---|---|---|---|
| skin<br>Assessment | ııme<br>Point | Statistic | M207<br>3.8 mg<br>(Sled) | M207<br>3.8 mg<br>(MACAP) | M207<br>3.8 mg<br>(MiniMac) |
| Erythema | Day 1, | | × × × | × > | ************************************** |
| | Fredose | SD | X.XX | XXXX | XX.X |
| | | Minimum | XX | XX | XX |
| | | Median | x.x | х.х | x.x |
| | | Maximum | XX | XX | XX |
| | Day 1, | и | × | × | × |
| | 30 Min | Mean | ×.× | x.x | ×× |
| | | SD | X.XX | X.XX | X.XX |
| | | Minimum | XX | XX | XX |
| | | Median | ×.× | x.x | x.x |
| | | Maximum | XX | XX | XX |

<Similar for all skin assessments and time points>

- made on a M207 3.8 mg (Sled): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application)

"Sled" coater and packaged in foil pouches (Treatment A)
M207 3.8 mg (MACAP): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made on a "MACAP" coater and packaged in foil cups (Treatment B)
M207 3.8 mg (MiniMac): M207 3.8 mg administered as two 1.9 mg patches 30 min wear time (upper arm application) - made

on a "MiniMac" coater and packaged in foil cups (Treatment

At each treatment and time point, the worst assessment scale between the two dosing patches application sites was used in the summaries. \* Scale descriptions:

Erythema: 0 = None; 1 = Mild redness; 2 = Moderate colored redness; 3 = Beet colored redness Edema: 0 = None; 1 = Slight edema; 2 = Moderate edema; 3 = Severe edema Bruising (visual rating): 0 = None; 1 =  $\leq 25$ % application site has bruising spots; 2 =  $\geq 26$  to  $\leq 50$ % application site has bruising spots;

3 = > 50% application site has bruising spots
Bleeding: 0 = None; 1 = Pink color on skin; 2 = Visible blood drop; 3 = Active bleeding
Program: /CAXXXXX/sas\_prg/stsas/tab programname.sas DDWMMYYY HH:MM

### 11. LISTING SHELLS

The following listing shells provide a framework for the display of data from this study. The shells may change due to unforeseen circumstances. These shells may not be reflective of every aspect of this study, but are intended to show the general layout of the listings that will be presented and included in the final report. These listings will be generated off of the Celerion SDTM Tabulation Model 1.4 mapped in accordance with SDTM Implementation Guide 3.2. All listings will be presented in Courier New font size 9.

Zosano Pharma Corporation M207, CP-2019-002 Celerion, Clinical Study Report No. CA27752

Appendix 16.1.10.1 Clinical Laboratory Reference Ranges


| Laboratory Group | Test Name | Sex | Age Category | Reference<br>Range | Units |
|---|---|---|---|---|---|
| Serum Chemistry | Test Name | XXXXXXX | XX | XX - XX | units |
| • | Test Name | XXXXXXX | × | × - × | units |
| | Test Name | XXXXXXX | XX | × - × | units |
| | Test Name | XXXXXXX | × | XX - XX | units |
| | Test Name | XXXXXXX | ×× | × - × | units |
| | Test Name | XXXXXX | × | XX - XX | units |
| Hematology | Test Name | XXXXXXX | × | XX - XX | units |
| · · | Test Name | XXXXXXX | × | | units |
| | Test Name | XXXXXXX | XX | | units |
| | Test Name | XXXXXXX | × | | units |
| | Test Name | XXXXXXX | × | | units |

<similar for remaining Laboratory Groups and Test Names>

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMMAME.sas DDMMMYYYY HH:NM

Appendix 16.2.1.1 Subject Discontinuation (All Randomized Subjects)


| ry Discontinuation<br>n | dverse Event |
|---|---|
| Primary I<br>Reason | Adver |
| Completed<br>Study? | YES<br>YES<br>NO |
| Date of<br>Completion or<br>Discontinuation | DDWWWIXXX<br>DDWWWIXXX<br>DDWWWIXXX |
| Actual<br>Treatment<br>Sequence | XXX |
| Randomized<br>Treatment<br>Sequence | XXX |
| Safety<br>Population | Yes<br>Yes<br>Yes |
| Subject<br>Number | ××× |

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMMANE.sas DDWAMYYYY HH:NM


Appendix 16.2.4.1 Demographics (Safety Population)

| Body Mass Informed<br>t Weight Index Consent<br>(kg) (kg/m²) Date | XX DDMMYYYY |
|---|---|
| Body Ma<br>Weight Index<br>(kg) (kg/m²) | xx.xx xx.xx |
| Height W | × |
| Ethnicity | Not Hispanic or Latino |
| Race | <b>^</b> |
| Sex | Male |
| Age*<br>(yrs) | X 2 |
| Date Of<br>Birth | DEMMMYYYY XX <similar above<="" td="" to=""></similar> |
| 44 | |

\* Age is derived from birth date to informed consent.

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMMAME.sas DDMMMYYYY HH:MM

Zosano Pharma Corporation M207, CP-2019-002 Celerion, Clinical Study Report No. CA27752

Appendix 16.2.4.2 Physical Examination Abnormal Findings (Safety Population)


| Description or Comment | ^ ^ ^<br>V V V |
|--------------------------------|--------------------------------------|
| System | XXXXX |
| Result | Abnormal<br>Abnormal<br>Abnormal |
| Date | DEMONYYYY<br>DEMONYYYY<br>DEMONYYYYY |
| Hour | XXX |
| -<br>Day | $\bowtie \bowtie$ |
| Treat-<br>ment | ×× |
| Study<br>Period | Screen<br>X<br>X |
| Subject Study<br>Number Period | × |

Treatment B: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >
HEENT = Head, Eyes, Ears, Nose, Throat

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DIMMMYYYY HH:NM

Zosano Pharma Corporation M207, CP-2019-002 Celerion, Clinical Study Report No. CA27752

Appendix 16.2.4.3 Medical and Surgical History (Safety Population)


| | | End Ongoing? Condition or Event | XX XXXXXXX XXXXXXXX XXXX | |
|---|---|---|---|---|
| | | | l | DDMMAXXX |
| Date | | Start | XXXXMMMXIQ<br>XXXXXMMMXIQ | TYYYYY |
| | | Category | XXXXX XXXXX Medical | Medical |
| | | Я | XXXXXX XXXXXX | XXXXXXXXXX |
| | Study | Period | Screen | Screen |
| | Anv | Number History? Period | X XXX Screen X | XXX |
| | Subject | Number | × | × |

Program: /CAXXXXX/sas\_prg/stsas/lis\_PRCGRAMMAME.sas DDMMMYYYY HH:NM

Appendix 16.2.4.4 Substance Use (Safety Population)


| End<br>Date | DDMMYYYY |
|-------------------------------------------------------------|--------------|
| Start End<br>Date Date | DDWWWYYY |
| Subject Study<br>Number Period Substance Description of Use | |
| Substance | XXX XXXXXXXX |
| Study<br>Period | Screen |
| Subject<br>Number | × |

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNEME.sas DDMMYYYY HH:NM

Appendix 16.2.5.1.1 Inclusion Criteria


\*\*\*\*

Appendix 16.2.5.1.2 Exclusion Criteria

\*\*\*\*\*\* \*\*\*\*\*\*

Program: /CAXXXXX/sas\_prg/stsas/lis\_programmame.sas DDWMMYYYY HH:MM

Appendix 16.2.5.2 Subject Eligibility (Safety Population)

| X Screen | X Screen | Subject Study Did<br>Number Period all eligi |
|---|---|---|
| YES | YES | subject m<br>bility cr |
| <pre><this are="" column="" data="" if="" is="" only="" present.="" presented=""></this></pre> | | eet<br>iteria? Specify |

Program: /CAXXXXX/sas\_prg/stsas/lis\_programmeme.sas DDMMYYYY HH:MM

Appendix 16.2.5.3 Check-in Responses (Safety Population)

| × | × | Number | Subject |
|---|---|---|---|
| × | × | Period | Study |
| × | × | ment | Treat- |
| $\stackrel{\ \ }{\ \ }\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!\!$ | × | Day | |
| XXXXX | XXXXX | Hour | |
| AAAAMMIIG | AAAAMMAID | Date | |
| HH:MM | MM:HH | Time | |
| Z Z | No | <br> | Check-in Criteria |
| <b>8</b> 8 | N | 2 | in Criteria* |
| there is a comment present in the study database. | Will only be present and populated if | Specify | |

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >
Treatm

Program: /CAXXXXX/sas\_prg/stsas/lis\_programmame.sas DDmmmyyyy HH:MM


Appendix 16.2.5.4 Test Compound Administration Times (Safety Population)

| ; | × | × | × | | Number | Subject | |
|---|---|---|---|---|---|---|---|
| ; | × | × | × | | Period | Study | |
| ż | ×; | | × | | ment | Treat- | |
| ÷ | × | | × | | Day | | |
| , | XXXX | | XXXX | | Hour | | |
| | ファインマンマン | TYYYMMICC | TYYYMMICC | | Date | the live had tracked in a large track and tracked track | Start |
| | ××××× | X:XX:XX | X:XX:XX | | Time | *************************************** | • |
| | XXXXXXXX | XXXXXXXXX | XXXXXXXXXX | | Compound | | |
| , | ^ ~ | ^<br>V | ^<br>V | *************************************** | Dosage | | |
| , | ^ ~ | ^ | ^ | | Laterality | | |
| , | ۸<br>٧ | ^<br>V | ^<br>V | | Form | | |
| , | ^ ^ | ^<br>V | ^<br>V | and the same arrange which and the same | Route | | |
| | | | XXXXXXXXXXXXXXXXXXXXXX | am am am pagang gang ang tagang tagang a tagang bank bank tank tank tank tank tank tank tank t | Comments | | |

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >
NA = Not applicable

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAWE.sas DDWWWYYYY HH:WM
Appendix 16.2.5.5 Blood Draw Times (Safety Population)

| | | | | | | 1 |
|---|---|---|---|---|---|---|
| | | | | | × | Subject<br>Number |
| | | | | | × | Study<br>Period |
| Simil: | | | | | × | Treat-<br>ment |
| lar for | × | × | × | × | × | Day |
| all other | XXXXXX | XXXXX | XXXXX | XXXXX | XXXXX | Hour |
| time point | XXXXMMMCO | AAAAMMADO | ALAKIMINGO | AAAAWWAAA | DDMMYYYY | Date |
| and subjec | HH:MM:SS XXX | HH:MM:SS | EH:IM:SS | HH:MM:SS | HH:MM:SS | Actual<br>Time |
| ቷs> | XXXXXXXX | XXXXXXXX | XXXXXXXXX | XXXXXXXX | XXXXXXXXX | Bioassay |
| | | | | | | Comments |
| | | | | | - 1 | |

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMMIME.sas DDMMMYYYY HH:MM

Appendix 16.2.5.6 Meal Times (Safety Population)

| Subject Study Treat- Number Period ment Day Hour Event Date Time Comments X X X XXXXX DINNER DDAMMYYYY XX:XX:XX XX:XX:XX X XXXXX SNACK DDAMMYYYY XX:XX:XX XX:XX:XX XXXXXX DINNER DDAMMYYYY XX:XX:XX XX:XX:XX XXXXXX DINNER DDAMMYYYY XX:XX:XX XX:XX:XX XXXXXX DINNER DDAMMYYYY XX:XX:XX XX:XX:XX XXXXXX DINNER DDAMMYYYY XX:XX:XX XX:XX:XX XXXXXX SNACK DDAMMYYYY XX:XX:XX XX:XX:XX XXXXXX XX:XX:XX XXXXXX SNACK DDAMMYYYY XX:XX:XX XXXXXX XX:XX:XX XXXXXX XX:XX:XX XXXXXX XX:XX:XX XXXXXX XX:XX:XX XXXXXX XX:XX:XX |
|---|
| Treat- ment Day Hour Event Date Time Time C X |
| - Day Hour Event Date Time C -X XXXXX DINNER DIMMYYYY XX:XX:XX XX:XX:XX X XXXXX SNACK DIMMYYYY XX:XX:XX XX:XX:XX X XXXXX DINNER DIMMYYYY XX:XX:XX XX:XX:XX X XXXXX DINNER DIMMYYYY XX:XX:XX XX:XX:XX XXXXX DINNER DIMMYYYY XX:XX:XX XX:XX:XX XXXXX DINNER DIMMYYYY XX:XX:XX XX:XX:XX XXXXX SNACK DIMMYYYY XX:XX:XX XX:XX:XX XXXXXX SNACK DIMMYYYY XX:XX:XX XX:XX:XX |
| Hour Event Date Time C XXXXX SUPCK DDMMYYYY XX:XX:XX XX:XX:XX XXXXX BREAKFAST DDMMYYYYY XX:XX:XX XX:XX:XX XXXXX DDNNER DDMMYYYYY XX:XX:XX XX:XX:XX XXXXX DDNNER DDMMYYYYY XX:XX:XX XX:XX:XX XXXXX DDNNER DDMMYYYYY XX:XX:XX XX:XX:XX XXXXX SUPCK DDMMYYYYY XX:XX:XX XX:XX:XX |
| Event Date Time C Event Date Time C X DINNER DDMMYYYY XX:XX:XX XX:XX:XX X SUNCK DDMMMYYYY XX:XX:XX XX:XX:XX X BREAKFAST DDMMMYYYY XX:XX:XX XX:XX:XX X DINNER DDMMYYYY XX:XX:XX XX:XX:XX X DINNER DDMMYYYY XX:XX:XX XX:XX:XX X SUNCK DDMMYYYY XX:XX:XX XX:XX:XX |
| Actual Start Stop Date Time Time C DDMMMYYYY XX:XX:XX XX:XX:XX |
| Start Stop Time Time C XX:XX:XX |
| Stop Time C XX:XX:XX C XX:XX:XX C XX:XX:XX C XX:XX:XX C XX:XX:XX C XX:XX:XX |
| ^^^^ |
| Comments |

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDXAMYYYY HH:NM

## Appendix 16.2.5.7 Prior and Concomitant Medications (Safety Population)

| | | | | 1 |
|---|---|---|---|---|
| | ω | 12 | ш | Subject |
| | YES | Ö | NO | t Any<br>Med? |
| × | | | | Treat-<br>ment |
| PARACETAMOL (PARACETAMOL) | (CETTRIZINE) | None | None | Treat- Medication<br>ment (WHO DD*) |
| × MG | × MG | | | Dosage |
| XXXXXXXXXX | HIDOM AE | | | Route |
| AAAAMMIGG | XXXXMMUU | | | Start |
| MW:HH | UNIK | | | Start<br>Time |
| HH:MM DDWMMYYYY HH:MM XXXXX | DDMMYYYY HH:MM XXXXXXX | | | Stop<br>Date |
| HH:MM | MW:HH | | | Stop |
| XXXXXXXX | XXXXXXX | | | Frequency |
| XXXXXXXXX | XXXXXXX | | ŀ | Indication |
| × | NO | | 77 | Prior<br>to<br>mency Indication Continuing? Study? |
| | Yes | | | Prior<br>to<br>Study? |

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >
\*Treatment D: < >
\*Concomitant medications are coded with WHO Dictionary Version OlMar2019-b3.
\*Med = Medication, UNK = Unknown, WHO DD = World Health Organization Drug Dictionary

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMMAME.sas DDMAMMYYYY HH:NM

Page 1 of X Appendix 16.2.6.3 Residual Amounts of Zolmitriptan in M207 Patches for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes in Healthy Volunteers (Safety Population)

| | | | | × | Subject<br>Number |
|-----------|----------|-----------|-----------|----------|-------------------|
| | | | | × | Study<br>Period |
| | | | | × | Treat-<br>ment |
| × | × | × | × | × | Day |
| XXXXX | XXXXX | XXXXX | XXXXX | XXXXX | Hour |
| AAAAMMICC | XXXXWWCD | XXXXWWXZQ | XXXXMMIDD | AAAAMWAA | Date |
| HH:MM:SS | HH:MM:SS | HH:MM:SS | HH:MM:SS | HH:MM:SS | Actual<br>Time |
| XXX | XXX | XXX | XXX | XXX | Result (µg) |

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMME.sas DIMMMYYYY HH:NM

Page 1 of X Appendix 16.2.6.4 Residual Amounts of Zolmitriptan on Skin Swabs for 3 Different Formulations of M207 3.8 mg on the Upper Arm for 30 Minutes in Healthy Volunteers (Safety Population)

| | } |
|--------------------------------------------------|-------------------|
| × | Subject<br>Number |
| × | Study<br>Period |
| × | Treat-<br>ment |
| **** | Day |
| XXXXX<br>XXXXX<br>XXXXX<br>XXXXX | Hour |
| XXXXWWCCC<br>XXXXWWCCC<br>XXXXWWCCC<br>XXXXWWCCC | Date |
| HH:MM:SS<br>HH:MM:SS<br>HH:MM:SS<br>HH:MM:SS | Actual<br>Time |
| XXX<br>XXX<br>XXX<br>XXX | Result (µg) |

Program: /CAXXXXX/sas\_prg/stsas/lis\_programMTME.sas DDMMMYYYY HH:MM

## Appendix 16.2.7.1.1 Adverse Events (I of II) (Safety Population)


| | ω | ω | 1 | Number | ?<br><br>)<br>} | |
|---|---|---|---|---|---|---|
| × | | | | Treatment | | |
| Yes | Ö | | | TE? | | |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXXXXXX | None | None | TE? Adverse Event | | 1 |
| XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | XXXXXXXXX/ XXXXXXXXX | | | Preferred Term* | Grater Owen Class | |
| <similar above="" to=""></similar> | DD:HH:MM | | | (DD:HH:MM) | Time From<br>Last Dose | |
| to above> | MW:HH XXXXMMOO | | | Date | Onset | |
| | HH:MM | | | Time | řŤ | |
| | WW:HH XXXXWWQQ | | | Date Time | Resolved | |
| | MY:HE | | | Time | Ď. | |
| | DD:HH:MM | | | (DD:HH:MM) | Duration | |

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >
Treatment D: < >
Treatment D: < >
\* Adverse events are coded using MedDRA Version 20.1.
TE = Treatment-emergent

Program: /CHXXXXX/sas\_prg/stsas/lis\_PROGRAMMAME.sas DIMMMYYYY HH:NM

Appendix 16.2.7.1.2 Adverse Events (II of II) (Safety Population)

| Treatment A: < > Treatment B: < > Treatment C: < > Treatment D: < > Serious: NS = Not Frequency: SE = Si | | Num | ടയം |
|---|---|---|---|
| ent A:<br>ent B:<br>ent C:<br>ent D:<br>: NS == | × | x I | ject |
| Treatment A: < > Treatment B: < > Treatment C: < > Treatment D: < > Serious: NS = Not Serious Frequency: SE = Single Ep | × | Number Treatment | |
| ous<br>Episode, | XXXXXXXXXX | Event | Adverse |
| Inter. = 1 | XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | | |
| Intermitte | DDA全全 | Date | |
| mt, Co | X XXXX | ļ | Onset |
| mt. = | X:XX | Time | 11 |
| Treatment A: < > Treatment B: < > Treatment C: < > Treatment D: < > Serious: NS = Not Serious Frequency: SE = Single Episode, Inter. = Intermittent, Cont. = Continuous | DRMMYYYY XX:XX Inter. | Frequency Severity Serious Outcome | |
| | Mild | Severity | |
| | NS | Serious | |
| | Recovered/<br>Resolved | | |
| | Recovered/XXXXXXXXX None<br>Resolved | Drug | Relation—<br>ship to<br>Study |
| | None | Action | |

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMMAME.sas DDMMMYYYY HH:MM

Appendix 16.2.7.2 Adverse Event Non-Drug Therapy (Safety Population)


| × | Subject<br>Number |
|---|---|
| X | Treatment |
| X X <> DDMMYYYY HH:MM DDMMYYYY HH:MM TRENDELENBURG POSITION | Adverse Event |
| MI:HH XXXXMMQQ | Onset<br>Date Time |
| WN:HH XXXXWWDD | Procedure Given Date Time Des |
| TRENDELENBURG<br>POSITION | Procedure Given Date Time Description |

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMMAME.sas DDMMMYYYY HH:NM

## Celerion, Clinical Study Report No. CA27752 Appendices 16.2.8.1.1 to 16.2.8.1.4 will be in the following format:

Appendix 16.2.8.1.1 Clinical Laboratory Report - Serum Chemistry (Safety Population)


| × | Subject<br>Number |
|----------------------------------------|----------------------------------|
| × | Age#/<br>Sex |
| Screen<br>X | Study<br>Period |
| ፟. | Day |
| ZZZZMMWOO | Date |
| SS:WW:HH A | Time |
| S XX EYR+ | Parameter1<br>< Range><br>(Unit) |
| XX<br>XX | Parameter2<br>< Range><br>(Unit) |
| ×× | Parameter3<br>< Range><br>(Unit) |
| -X1 XX<br>XX | Parameter4<br>< Range><br>(Unit) |
| XX | Parameter5<br>< Range><br>(Unit) |
| ×× | Parameter6 < Range> (Unit) |

# Age is derived from birth date to date of informed consent. F = Female, M = Male H = Above reference range, L = Below reference range

Computer: N = Not clinically significant, Y = Clinically significant

PI Interpretation: - = Not clinically significant, R = Recheck requested, ^ = Will be retested later, + = Clinically significant

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNAME.sas DDMMMYYYY HH:MM

Programmer Note: Replace Parameter1, 2 etc. with actual lab tests in the study. Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for.

Add fourth flag in the cases that ^ or R are used for the PI flag. This flag will be found in the ClinQuick Extraction.

Appendix 16.2.8.1.5 Clinical Laboratory Report - Comments (Safety Population)

| × | Number |
|---|---|
| × | Sex |
| × | Period |
| × | Day |
| AXXAMMIGG | Number Sex Period Day Date |
| DDWWYYYY Other Tests | Department |
| Fibrinogen | Number Sex Period Day Date Department Test Result Unit Con |
| XXX | Result |
| mg/dL | Unit |
| Not significant in the context of this study. | Connent |

# Age is derived from birth date to date of informed consent. F = Female, M = Male

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMMPME.sas DDMMMYYYY HH:NM


Appendix 16.2.8.2 Vital Signs (Safety Population)

| × | Subject<br>Number |
|---|---|
| XCreen | |
| ×× | Treat-<br>ment |
| ××· | Day |
| ××. | Hour |
| XXXXVVVCC<br>XXXXVVVCC<br>XXXXVVVCC | Date |
| X | Time |
| XEIIX | Bloc<br>Test |
| XXX/ XX<br>XXX/ XX | Blood Pressure (mmHg) Test Systolic/Diastolic |
| *** | (bpm) |
| ××× | Respi-<br>ration<br>(bpm) |
| × | Tempera-<br>ture<br>(°C) |
| XXX.<br>.x | espi- Tempera-<br>stion ture Weight<br>gm) (°C) (kg) Comment |
| | Comment |

**Programmer Note:** Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for.

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >
For pulse, bpm is beats/minute and for respiration bpm is breaths/minute.
SITX = X-minute sitting, SUPX = X-minute supine, R = Recheck value

Program: /CAXXXXX/sas\_prg/stsas/lis\_PROGRAMNUME.sas DDMMYYYY HH:1MM


Appendix 16.2.8.3 12-Lead Electrocardiogram (Safety Population)

| × | Subject<br>Number |
|----------------------------------------|------------------------|
| | ject<br>ber |
| Screen<br>X | Study |
| × | Treat-<br>ment |
| ×· | _<br>Day |
| XXX. | Hour |
| XXXXMMDD | Date |
| X:XX:XX | Time |
| Normal<br>Normal | Result |
| ×× | Heart<br>Rate<br>(bpm) |
| XXX.X | PR<br>(ms) |
| ×.× | QRS<br>(ms) |
| XXX.X | (mg) |
| XXX.X | QTcF*<br>(ms) |
| X.XXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXXX | Comment |

**Programmer Note:** Sort unscheduled assessment and early term chronologically with other scheduled assessments and rechecks. Recheck should be sorted with the scheduled time point the recheck is for.

Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >
QTcF\* = QT corrected for heart rate using Fridericia's correction
# = QTc >= 450 ms, @ = QTc change from baseline greater than or equals to 30 ms.

Program: /CAXXXXX/sas\_prg/stsas/lis\_programmame.sas MW:HH XXXXMMUD


Appendix 16.2.8.4 Investigator Visual Skin Assessments (Safety Population)

| | 19 A | n |
|---|---|---|
| × | Jumber<br>Jecc | Subject |
| XXXX X X XXXX | Number Period | C<br>t |
| × | Treat-<br>ment Day | |
| ×× | Day | 1 |
| XXX | Hour | |
| XXXXMMIGG<br>XXXXMMIGG | Da⊤e | |
| X:XX | Time | |
| ×× | Erythema | |
| ×× | Edema | Skin A |
| ×× | Bruising | Skin Assessment* |
| ×× | Erythema Edema Bruising Bleeding | |
| XXXXXXXXXXXXXXXXX | Comments | |

```
Treatment A: < >
Treatment B: < >
Treatment C: < >
Treatment D: < >
Erythema: 0 = None; 1 = Mild redness; 2 = Moderate colored redness; 3 = Beet colored redness

Edema: 0 = None; 1 = Slight edema; 2 = Moderate edema; 3 = Severe edema

Edema: 0 = None; 1 = Slight edema; 2 = Moderate edema; 3 = Severe edema

Bruising (visual rating): 0 = None; 1 = ≤ 25% application site has bruising spots; 2 = ≥ 26 to ≤ 50% application site has bruising spots; 3 = > 50% application site has bruising spots

Bleeding: 0 = None; 1 = Pink color on skin; 2 = Visible blood drop; 3 = Active bleeding
                                                                                                                                                                                                                                                                                  * Scale descriptions:
```

Program: /CAXXXXX/sas\_prg/stsas/lis\_programwame.sas DDMMYYYY HH:MM

| • |
|---|

.